## Statistical Analysis Plan J1V-MC-BT01 Version 3

A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Two-Arm, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of LY3361237 as a Treatment for Adults With At Least Moderately Active Systemic Lupus Erythematosus.

NCT05123586

Approval Date: 31-Aug-2023

# Statistical Analysis Plan:

# J1P-MC-BT01: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3361237 as a Treatment for Adults with At Least Moderately Active Systemic Lupus Erythematosus

**Master Protocol Title:** A Master Protocol for a Randomized, Placebo-Controlled Clinical Trial of Multiple Interventions for the Treatment of Systemic Lupus Erythematosus

Master Protocol Number: J1V-MC-IMMA Master Compound Number: LY900024

Master Protocol Short Title: A Master Protocol for a Randomized, Placebo-Controlled Clinical

Trial of Multiple Interventions for the Treatment of Systemic Lupus Erythematosus

Sponsor Name: Eli Lilly and Company

Legal Registered Address: Eli Lilly and Company, Indianapolis, Indiana, USA 46285

Regulatory Agency Identifier Number(s)

IND: 155806

### List of Intervention-Specific Appendices (ISAs):

ISA 1 for LY3361237 versus placebo (J1V-MC-BT01)

**ISA Title:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Two-Arm, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of LY3361237 as a Treatment for Adults with At Least Moderately Active Systemic Lupus Erythematosus

ISA Number: J1V-MC-BT01

ISA Compound Number: LY3361237

Study Phase: 2

**ISA Short Title:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Two-Arm, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of LY3361237 to Treat Adults with At Least Moderately Active Systemic Lupus Erythematosus

### Confidential Information

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiaries

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

**Document ID: VV-CLIN-117498** 

# **Table of Contents**

| Secti | on | Page |
|---|---|---|
| Statis | tical Analysis Plan: J1P-MC-BT01: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Study of LY3361237 as a Treatment for Adults with At Least Moderately Active Systemic Lupus | |
| 115 | Erythematosus | |
| 1. | Introduction | |
| 1.1. | Objectives and Estimands | |
| 1.2. | Study Design | |
| 2. | Statistical Hypotheses | |
| 2.1. | Multiplicity Adjustment | 12 |
| 3. | Analysis Sets | 13 |
| 4. | Statistical Analyses | 14 |
| 4.1. | General Considerations | |
| 4.2. | Participant Characteristics | 16 |
| 4.2.1. | Demographics and Baseline Characteristics | |
| 4.3. | Participant Disposition | 16 |
| 4.4. | Primary Estimand. | 16 |
| 4.4.1. | Main Analytical Approach. | 17 |
| 4.4.1.1 | | |
| 4.5. | Secondary Estimand(s) | |
| 4.5.1. | Additional Analysis | |
| 1.6. | Supplementary Estimands for Primary and Secondary Objectives | |
| 4.7. | Exploratory Estimands | |
| 4.7.1. | Rash and Arthritis | 20 |
| 4.7.2. | Rash and/or Arthritis with Intercurrent Events Handled Using Treatment | - Marie 1 |
| | Policy Strategy | |
| 4.7.3. | Corticosteroid-Sparing Effect | 21 |
| 4.7.4. | Individual Organ System Systemic Lupus Erythematosus Disease | |
| | Manifestations Using Systemic Lupus Erythematosus Disease Activity | |
| | Index 2000 Components, Cutaneous Lupus Erythematosus Disease Area and Severity Index, and Joint Counts | 21 |
| 4.7.5. | Lupus Low Disease Activity State | |
| 4.7.6. | British Isles Lupus Assessment Group-Based Composite Lupus | 22 |
| 4.7.0. | Assessment | 23 |
| 4.7.7. | Physician's Global Assessment of Disease Activity | |
| 4.7.8. | Time to, and Incidence of, Any Flare and First Severe Flare | |
| 4.7.9. | Serologic Markers of Systemic Lupus Erythematosus | |
| 4.7.10 | | |
| 4.7.11 | . Systemic Lupus Erythematosus International Collaborating Clinics | |
| | Damage Index | 24 |
| 4.8. | Safety Analyses | 24 |
| 4.8.1. | Extent of Exposure. | |
| 4.8.2. | Adverse Events | 26 |

| 4.8.2.1 | . Adverse Events | 26 |
|---|---|---|
| 4.8.2.2 | Serious Adverse Events | 27 |
| 4.8.3. | Adverse Events of Special Interest | 28 |
| 4.8.3.1 | | |
| 4.8.3.2 | | |
| 4.8.4. | Injection Site Reaction | |
| 4.8.5. | Clinical Laboratory Evaluations | 31 |
| 4.8.6. | Vital Signs and Other Physical Findings | 31 |
| 4.8.7. | Depression and Suicide | 31 |
| 4.9. | Other Analyses | 32 |
| 4.9.1. | Concomitant Therapy | 32 |
| 4.9.2. | Treatment Compliance | 32 |
| 4.9.3. | Immunogenicity Assessments | 32 |
| 4.9.4. | Patient-Reported Outcomes | 33 |
| 4.9.5. | Subgroup Analyses | 33 |
| 4.10. | CCI | 34 |
| 4.10.1. | Assessment Committee | 34 |
| 4.11. | Pharmacokinetic Assessment | 35 |
| 4.12. | Pharmacodynamic Assessment | 35 |
| 4.13. | Data Monitoring Committee | 35 |
| 4.14. | Changes to Protocol-Planned Analyses | 35 |
| 5. | Sample Size Determination | 36 |
| 6. | Supporting Documentation | 37 |
| 6.1. | Appendix 1: Description and Derivation of Efficacy Outcomes Measures | |
| | and Endpoints | 37 |
| 6.2. | Appendix 2: Description of Efficacy Analyses | 44 |
| 6.3. | Appendix 3: SLEDAI-2K | |
| 6.4. | Appendix 4: BILAG 2004 | |
| 6.5. | Appendix 5: Joint Assessment | |
| 6.6. | Appendix 6: SLICC/ARC Damage Index | 66 |
| 6.7. | Appendix 7: Corticosteroid Conversion | 66 |
| 6.8. | Appendix 8: Corticosteroid Management | 68 |
| 6.9. | Appendix 9: List of MedDRA Preferred Terms for Potential Opportunistic | |
| | Infections | 69 |
| 6.10. | Appendix 10: List of Planned Laboratory Analytes with Reference Range | |
| | Sources | 83 |
| 6.11. | Appendix 11: Common Terminology Criteria for Adverse Events Related | |
| | to Myelosuppressive Events | 87 |

# **Table of Contents**

| Table | | Page |
|------------|--------------------------------------|------|
| Table 1. | SAP Version History Summary | 6 |
| Table 4.1. | ISA Specific Patient Characteristics | 16 |

# **Table of Contents**

| Figure | | Page |
|---|---|---|
| Figure 1. | Schema of Study J1V-MC-BT01, a Phase 2 study to evaluate the efficacy and safety of LY3361237 in adults with at least moderately active systemic lupus erythematosus. | 10 |

# **Version History**

This statistical analysis plan (SAP) for Study J1V-MC-BT01 (BT01) is based on the protocol dated 22 September 2021.

Study BT01 SAP version 3 was approved prior to the unblinding for a planned interim analysis of the first ISA (Study BT01). Changes in version 3 are documented. Minor corrections and/or additions may not be included.

Table 1. SAP Version History Summary

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|---|---|---|---|
| 1 | 9 Feb 2022 | Not Applicable | Original version |
| 2 | 15 Feb 2022 | Update Table of<br>Contents and<br>minor editing | New comments in the SAP, link sections in the document |
| 3 | See date on<br>Page 1 | Update Sections<br>1, 4, and 6 and<br>minor edits | Align with the analysis in previous studies and new comments |

### 1. Introduction

This statistical analysis plan (SAP) is for Study J1V-MC-BT01 (BT01), an intervention-specific appendix (ISA) to the Master Protocol J1V-MC-IMMA (IMMA). This SAP has been developed after review of the Study BT01 Clinical Study Protocol (final version dated 21 June 2021), and Study BT01 Protocol Amendment (a) (final version dated 22 September 2021).

This SAP describes the planned analysis of the efficacy, safety, and pharmacokinetic (PK) and pharmacodynamic (PD) data from this study. A detailed description of the planned tables, figures, and listings (TFLs) to be presented in the clinical study report (CSR) is provided in the accompanying TFL shell document.

The intent of this document is to provide guidance for the statistical, PK and PD analyses of data. In general, the analyses are based on information from the protocol and there are no changes to the analyses described in the protocol. A limited amount of information concerning this study (for example, objectives, study design) is given to help the reader's interpretation. When the SAP and TFL shells are agreed upon and finalized, they will serve as the template for this study's CSR.

SAP BT01 elaborates on the statistical considerations identified in Protocol BT01 and SAP BT01 cannot modify the primary and secondary analyses described in Protocol BT01. If additional analyses are required to supplement the planned analyses described in SAP BT01, then these analyses may be performed and will be identified in each ISA's clinical study report (CSR) as post hoc analyses. Any minor deviations from the TFLs may not be documented in the CSR.

This SAP is written with consideration of the recommendations outlined in the International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials<sup>1</sup> and the ICH E3 Guideline entitled Guidance for Industry: Structure and Content of Clinical Study Reports<sup>2</sup>.

# 1.1. Objectives and Estimands

| Objectives | Estimands |
|---|---|
| Primary | |
| To compare the efficacy of 450 mg LY3361237 Q2W versus placebo with respect to arthritis and/or rash remission in participants with SLE | The study will compare LY3361237 Q2W with placebo as randomized in participants with moderate to severe SLE who present with arthritis and/or rash at baseline. |
| | The primary comparison is the difference in proportions of participants who |
| | <ul> <li>achieve remission of arthritis and/or rash as defined by SLEDAI-2K at Week 24</li> <li>do not discontinue from treatment for any reason, and</li> <li>do not violate concomitant medication rules.</li> </ul> |
| Secondary | |
| To compare 450 mg LY3361237 Q2W versus placebo with respect to SLE clinical signs and symptoms treatment response | The study will compare LY3361237 Q2W with placebo as randomized in participants with moderate to severe SLE who present with arthritis and/or rash at baseline. |
| | <ul> <li>difference in proportions of participants who achieve SLEDAI-4 response at Week 24 and do not discontinue from treatment for any reason and not violate commitment medication rules, and</li> <li>difference in proportions of participants who achieve SRI-4 response at Week 24 and do not discontinue from treatment for any reason and not violate commitment medication rules.</li> </ul> |

| • | To characterize the PK of 450 mg |
|---|------------------------------------|
| | LY3361237 Q2W in participants with |
| | SLE |

Steady-state trough serum concentration of LY3361237 at Week 24

### **Exploratory Objectives**

The following are exploratory objectives for the evaluation of 450 mg LY3361237 Q2W:

- To compare the efficacy of LY3361237 Q2W versus placebo for the following measures:
  - o corticosteroid sparing effect
  - o individual organ system SLE disease manifestations using
    - SLEDAI-2K components
    - CLASI, and
    - joint counts
  - o measures of SLEDAI-2K low-disease activity
    - LLDAS
  - o BICLA
  - o PGA
  - o time to, and incidence of, any flare and first severe flare
  - o serologic markers of SLE
  - o interferon gene signature, and
  - o SLICC/ACR Damage Index.
- To describe the observed safety of LY3361237 Q2W.
- To assess the potential development of anti-LY3361237 antibodies.
- To characterize the exposure-response of LY3361237 Q2W as related to biomarkers, RO, efficacy, and safety endpoints.
- To explore the effect of LY3361237 Q2W on exploratory biomarkers of SLE disease activity.

**Note:** The precise analysis for each estimand will be prospectively defined in the following sections of the statistical analysis plan and will include, at minimum, drug to be evaluated, dose/dosing regimen, population, indication under study, comparator, and timing of the analysis.

Abbreviations: ACR = American College of Rheumatology; BICLA = BILAG-based Composite Lupus Assessment; BILAG = British Isles Lupus Assessment Group; CLASI = Cutaneous Lupus Erythematosus Disease Area and Severity Index; LLDAS = lupus low disease activity state; PGA = Physician's Global Assessment of Disease Activity; PK = pharmacokinetics; Q2W = every 2 weeks; RO = receptor occupancy; SLE = systemic lupus erythematosus; SLEDAI-2K = Systemic Lupus Erythematosus Disease Activity Index 2000; SLEDAI-4 = defined as a ≥4-point reduction in SLEDAI-2K score from baseline; SLICC = Systemic Lupus Erythematosus International Collaborating Clinics; SRI-4 = Systemic Lupus Erythematosus Responder Index-4.

### 1.2. Study Design

Study BT01 is an ISA to Master Protocol IMMA. It is a multinational, multicenter, randomized, double-blind, placebo-controlled, parallel-group, 2-arm Phase 2 study to evaluate the efficacy and safety of LY3361237 plus standard of care in adult study participants with at least moderately active systemic lupus erythematosus (SLE). This ISA has a required treatment period and a required post-treatment follow-up period. Master Protocol IMMA describes an optional prescreening period and a required screening period.

### **Number of Participants:**

Approximately 90 participants will be randomly assigned in a 1:1 ratio to either LY3361237 or placebo. A schematic of the overall study design is presented in Figure 1.



Abbreviations: FD = first dose; ISA = intervention-specific appendix; LD = last dose; R = randomization to intervention groups of ISA; V = visit; W = week.

Figure 1. Schema of Study J1V-MC-BT01, a Phase 2 study to evaluate the efficacy and safety of LY3361237 in adults with at least moderately active systemic lupus erythematosus.

### Optional prescreening period

The optional prescreening period is described in the Study IMMA SAP (Section 1.2.1).

### Screening period

The screening period is described in the Study IMMA SAP (Section 1.2.1). The ISA specific informed consent forms will be signed before any Visit 2 study procedures are performed.

Participants found to be eligible according to all the study entry criteria of both Master Protocol IMMA and this ISA will be randomly assigned in a 1:1 ratio to receive 1 of the following study interventions:

- 450 mg LY3361237 once every 2 weeks (Q2W) plus standard of care, and
- placebo plus standard of care, given at matching intervals.

Participants will be stratified at randomization according to disease activity at baseline, corticosteroid dose at baseline, and geographic region (See Section 6.3 of Protocol BT01). Study interventions will be administered by subcutaneous (SC) injection.

### Double-blind treatment period

Randomized participants will begin the double-blind, placebo-controlled, 24-week treatment period at Visit 2. Participants will receive the first dose of the assigned study intervention at that visit and will continue to receive doses through the last scheduled dosing visit specified in the Schedule of Activities (Section 1.3 of Protocol BT01). Participants will maintain their usual standard of care medication regimen for SLE and for other diseases throughout the study, unless these medication regimens are specifically excluded (see Sections 5.2 and 6.5 of the Master Protocol IMMA) or unless changes are explicitly required by this Protocol BT01 (for example, dose adjustment for corticosteroids [see Section 6.5.1]). Safety and efficacy assessments and laboratory sample collections will be performed as specified in the Schedule of Activities (Section 1.3 of Protocol BT01) and as described in the Master Protocol IMMA.

### Follow-up period

The posttreatment follow-up visit lasts approximately 10 weeks after the last visit of the 24-week treatment period. All participants will have posttreatment follow-up visits (Visit 801 and Visit 802; see Section 1.3 of Protocol BT01) for sample collections, including anti-drug antibodies (ADA) and PK, and for safety assessments.

### Early discontinuation of study intervention

Participants who permanently discontinue the study intervention early are encouraged to remain in the study for safety monitoring through the end of the study treatment period and to participate in posttreatment follow-up visits. See Section 7 of the Master Protocol IMMA.

### 2. Statistical Hypotheses

The primary objective is to compare LY3361237 to placebo regarding remission of arthritis and/or rash at Week 24. Thus, the null hypothesis to be tested in relation to the primary estimand is as follows:

• Null hypothesis: LY3361237 is not different from placebo with respect to the achievement of remission of arthritis and/or rash at Week 24.

The null hypotheses corresponding to the secondary estimands are as follows:

- LY3361237 is not different from placebo with respect to the achievement of Systemic Lupus Erythematosus Responder Index-4 (SRI-4) at Week 24, and
- LY3361237 is not different from placebo with respect to the achievement of a ≥4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score from baseline (SLEDAI-4) at Week 24.

Additionally, we will test some exploratory hypotheses for arthritis and rash respectively:

- Null hypothesis: LY3361237 is not different from placebo with respect to the change of arthritis status (improvement, no change, worsening) at Week 24, and
- Null hypothesis: LY3361237 is not different from placebo with respect to the change of rash status (improvement, no change, worsening) at Week 24.

### 2.1. Multiplicity Adjustment

No adjustments for multiplicity will be performed.

### 3. Analysis Sets

For the purposes of analysis, the following analysis sets are defined.

| Participant Analysis Set | Description |
|---|---|
| Full analysis set | <ul> <li>All randomized participants. Participants will be included in the analyses<br/>according to the planned intervention.</li> </ul> |
| mITT analysis set | <ul> <li>All participants randomly assigned to study intervention and who take at<br/>least 1 dose of study intervention. Participants will be included in the<br/>analysis set according to their randomly assigned intervention.</li> </ul> |
| BICLA analysis set | <ul> <li>All mITT participants who meet the eligibility criteria for BICLA<br/>assessment. The eligibility criteria detail is in Section 4.7.6.</li> </ul> |
| PP analysis set | All randomized patients who do not commit an IPD that could potentially compromise efficacy results. IPDs are specified in the Trial Issue Management Plan. |
| Biomarker evaluable analysis set | <ul> <li>All randomized patients within the subset of participants from the<br/>exploratory analyses of dose and/or exposure relationship from whom a<br/>valid assay result has been obtained.</li> </ul> |
| Safety analysis set | <ul> <li>All participants randomly assigned to study intervention and who take at<br/>least 1 dose of study intervention. Participants will be analyzed according<br/>to the intervention they actually received within each study period.</li> </ul> |
| PK/PD analysis set | <ul> <li>All participants receiving at least 1 dose of study intervention and have<br/>PK and RO data available.</li> </ul> |

Abbreviations: BICLA = BILAG-based Composite Lupus Assessment; BILAG = British Isles Lupus Assessment Group; IPD = Important Protocol Deviation; mITT = modified intent-to-treat; PD = pharmacodynamic; PK = pharmacokinetic; PP = per-protocol; RO = receptor occupancy.

The safety analysis set is used to analyze the endpoints and assessments related to safety, and the modified intent-to-treat (mITT) and the per-protocol (PP) populations will be used in analyses of efficacy and patient-reported outcomes (PRO), unless otherwise specified. All protocol deviations that occur during the study will be considered for their severity/impact and will be taken into consideration when participants are assigned to analysis populations.

### 4. Statistical Analyses

### 4.1. General Considerations

This SAP is intended to describe the analyses of all objectives, as well as safety assessments, for Study BT01.

Statistical analysis of this study will be the responsibility of Eli Lilly and Company or its designee. For primary and key secondary objectives, statistical analyses will be performed using SAS® Enterprise 7.1 or higher, or SAS® Version 9.4 or higher.

See Master Protocol IMMA (Section 9.3.1) and Master Study IMMA SAP for platform trial considerations, such as borrowing of placebo data.

Considerations specific to this ISA include the following:

- All efficacy analyses will be tested at a two-sided alpha level of .10 for frequentist analyses.
- The primary and secondary estimand that will be used to analyze the primary and secondary endpoints is composite strategy estimand where comparisons will not include data collected after intercurrent events (ICE) including any concomitant medication violation or treatment discontinuation. Participants who discontinue or who are noncompliant with concomitant medication rules are defined as non-responders. Endpoint definition effectively gives complete data which will be analyzed as described in Sections 4.4 and 4.5.
- The p-values will be rounded up to 3 decimal places. For example, any p-value strictly >.049 and ≤.05 will be displayed as .050. This guarantees that on any printed statistical output, the unrounded p-value will always be less than or equal to the displayed p-value. A displayed p-value of .001 will always be understood to mean ≤.001. Likewise, any p-value displayed as 1.000 will be understood to mean >.999 and ≤1.

Not all displays described in this SAP will necessarily be included in the CSR. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools such as Spotfire instead of, or in addition to, a static display. Any display described in this SAP and not included in the CSR would be available upon request.



The treatment response rates, treatment differences versus placebo, and their corresponding 90% CIs will be provided.

The primary analysis method for both unconditional treatment difference of continuous efficacy and health outcome variables will be G-computation using a linear regression model with treatment group (LY or placebo), baseline disease activity (SLEDAI-2K <10 or SLEDAI-2K ≥10), corticosteroid dose at baseline (<10 mg/day or ≥10 mg/day), geographic region (USA, Europe, or rest of the world) in the model. The mean for each treatment group along with the estimate of the difference between treatments (difference between LY group and placebo), standard error (SE), p-value, and the 90% CIs will be reported at each visit along with p-values. For variables that are not collected at each postbaseline visit, data may exist at visits where the variable was not scheduled to be collected, due to early discontinuation visits. In these situations, data from the early discontinuation visit that do not correspond to the planned collection schedule will be excluded from the linear regression analyses. However, the data will still be used in other analyses. In addition, if an ICE happens, including but not limited to rescue medication use, the data collected before that event will be used and any data afterward will be excluded in the linear regression model.

The Kaplan-Meier product limit method will be used to estimate the survival curves for time-to-event variables.

Treatment comparisons will

use the hazard ratios and corresponding p-values from the Cox regression. Patients completing the treatment period without event will be censored at the date of completion. Patients without an event, a date of completion, or discontinuation for the treatment period will be censored at the latest nonmissing date out of the following dates: date of last dose and date of last attended visit in the treatment period. Under the hypothetical estimand strategy, patients without an event prior to the first violation of concomitant medication rules will be censored at the time of the first violation of concomitant medication rules.

Descriptive statistics will be used to summarize for all adverse events (AE), discontinuation, and other categorical safety data. Continuous vital signs and laboratory values will be analyzed using descriptive summaries and may also by a linear regression model with treatment and baseline values in the model. Statistics to be presented are the same as those for linear regression analyses stated above. For document writing purposes for safety, tests with two-sided p-values less than .10 will be referred to as having significant statistical evidence for a treatment difference, unless otherwise noted.

Efficacy and PRO analysis models may contain the independent variables such as treatment group, baseline disease activity, and geographic region.

### Changes to the data analysis methods

SAP BT01 elaborates on the statistical analysis specified in Protocol BT01. Any change to the data analysis methods described in SAP BT01, and the justification for making the change, will be described in the CSR and should be considered post hoc, regardless of whether the change occurred before unblinding or not. Furthermore, additional exploratory analyses of the data will be conducted as deemed appropriate and will be considered post hoc.

### 4.2. Participant Characteristics

### 4.2.1. Demographics and Baseline Characteristics

Refer to Section 4.4.1 in Study IMMA SAP for summaries of participant demographics and baseline characteristics. Additional ISA specific analysis is described in Table 4.1.

Table 4.1. ISA Specific Patient Characteristics

| Variable | Continuous | Categorical Summary | Subgroup Analysis |
|---|---|---|---|
| Disease Severity at Baseline | | | |
| Total SLICC/ACR Damage Index score | Yes | None | |

Abbreviations: ACR = American College of Rheumatology; SLICC = Systemic Lupus International Collaborating Clinics.

### 4.3. Participant Disposition

Please refer to Section 4.5 of Study IMMA SAP for Participant Disposition.

### 4.4. Primary Estimand

### Remission of arthritis and/or rash at Week 24

The primary clinical question of interest is: What is the difference between LY3361237 and placebo in the target patient population, in the proportion of participants who achieve remission of arthritis and/or rash as defined by the SLEDAI-2K after 24 weeks of intervention without violating concomitant medication rules and do not discontinue study intervention?

The ICEs of interest – "intervention discontinuation for any reason" and "any concomitant medication violation" – will be handled through the endpoint definition (composite variable strategy) and will be considered non-responders. All remaining ICEs are handled using the treatment policy strategy.

The estimand is described by the following attributes:

**Population:** participants with moderate to severe SLE who present with arthritis and/or rash at baseline. Further details can be found in Protocol BT01 Section 5.

**Endpoint:** responders at Week 24 defined as achieving all 3 of the following criteria:

- achieves remission of arthritis and/or rash at Week 24 as measured by SLEDAI-2K and defined in Protocol BT01 Section 8.1.1
- · does not permanently discontinue study intervention for any reason prior to Week 24, and
- does not violate any concomitant medication rules (Protocol BT01 Section 6.5 and Section 6.8 of this SAP) prior to Week 24.

**Treatment condition:** study interventions as randomized with restricted use of concomitant medications. Further details on study interventions and concomitant medications can be found in Protocol BT01 Section 6.

**Population-level summary:** Unconditional difference in proportions of responders at Week 24 between treatment conditions (LY3361237 vs. placebo).

The rationale for this estimand is that if a participant discontinues treatment, the burden of treatment outweighs its benefits. It also assumes that if a participant violates the concomitant medication rules, the participant is not receiving sufficient benefit from treatment. Therefore, being a responder requires a positive response as well as completing treatment and not violating concomitant medication rules.

### 4.4.1. Main Analytical Approach

The primary endpoint analysis will use the mITT population. The primary endpoint will be analyzed using a G-computation with logistic regression model as working model to test the treatment difference between LY3361237 450 mg versus placebo in the proportion of patients who achieve remission of arthritis and/or rash at Week 24 with the stratification at randomization variables including the baseline disease activity, corticosteroid dose at baseline, and geographic region as model covariates.

The unconditional odds ratio and 90% CIs will be reported. The unconditional treatment difference and 90% CIs will be reported. In addition, we will report the 95% CIs and the p-values with respect to the alpha threshold .05.

### Stratification at randomization

The randomization will be stratified based on the following factors:

- disease activity at baseline (SLEDAI-2K <10; SLEDAI-2K ≥10)</li>
- corticosteroid dose at baseline (<10 mg; ≥10 mg), and</li>
- geographic region (United States; Europe; rest of the world).

### 4.4.1.1. Missing Data Imputation

| CCI |
|-----|

### CCI

### 4.5. Secondary Estimand(s)

### SLEDAI-4 at Week 24

The clinical question of interest for a secondary objective regarding reduction in other SLE clinical signs and symptoms is: What is the difference in the percentage of participants who achieve SLEDAI-4 after 24 weeks of intervention without violating concomitant medication rules and do not discontinue study intervention?

The same ICE strategies used for constructing the primary estimand will be used for constructing this estimand.

The estimand is described by the following attributes:

**Population:** participants with moderate to severe SLE who present with arthritis and/or rash at baseline. Further details can be found in Protocol BT01 Section 5.

**Endpoint:** responder at Week 24 defined as achieving all 3 of the following criteria:

- achieves SLEDAI-4 response at Week 24 as defined in the Protocol BT01 Section 8.1.2.1
- · does not permanently discontinue study intervention for any reason prior to Week 24, and
- does not violate any concomitant medication rules (Protocol BT01 Section 6.5 and Section 6.8 of this SAP) prior to Week 24.

**Treatment condition:** study interventions as randomized with restricted use of concomitant medications. Further details on study interventions and concomitant medications can be found in Protocol BT01 Section 6.

**Population-level summary:** unconditional difference in proportions of responders at Week 24 between treatment conditions (LY3361237 vs. placebo).

The rationale for this estimand is the same as the primary estimand.

#### SRI-4 at Week 24

The clinical question of interest for another secondary objective regarding reduction in other SLE clinical signs and symptoms is: What is the difference between the proportion of participants who achieve SRI-4 after 24 weeks of intervention without violating concomitant medication rules and do not discontinue study intervention?

The same ICE strategies used for constructing the primary estimand will be used for constructing this estimand.

The estimand is described by the following attributes:

**Population:** participants with moderate to severe SLE who present with arthritis and/or rash at baseline. Further details can be found in Protocol BT01 Section 5.

**Endpoint:** responder at Week 24 defined as achieving all 3 of the following criteria:

- achieves SRI-4 response at Week 24 as defined in Protocol BT01 Section 8.1.2.2.
- does not permanently discontinue study intervention for any reason prior to Week 24, and
- does not violate any concomitant medication rules (Protocol BT01 Section 6.5 and Section 6.8 of this SAP) prior to Week 24.

**Treatment condition:** study intervention as randomized with restricted use of concomitant medications. Further details on study interventions and concomitant medications can be found in Protocol BT01 Section 6.

**Population-level summary:** Unconditional difference in proportions of responders at Week 24 between treatment conditions (LY3361237 vs. placebo).

The rationale for this estimand is the same as the primary estimand. The missing data will be handled similarly to the process described in Section 4.4.1.1.

### 4.5.1. Additional Analysis

The number and percentage of responders and non-responders at each visit will be presented by treatment group. The proportion of responders to SRI-4 at treatment completion will be analyzed using a logistic regression model as specified for the primary analysis in Section 4.4.1. Moreover, the number and percentage of patients who sustain responses will be summarized by treatment group. Specifically, 1 type of sustained response will be included:

respond by Week 12 and maintain response until Week 24.

A table for reasons of non-response, based on NRI, will also be tabulated at Week 24. Reasons are study treatment non-completers, concomitant medication violation (increase), SLEDAI not reduced by ≥4 points, British Isles Lupus Assessment Group (BILAG) criteria not met, Physician's Global Assessment (PGA) criteria not met, or missing data. If a patient is a non-responder by more than 1 reason, then count only the first reason in the list. For example, if a patient didn't meet SLEDAI criteria and BILAG criteria, then the patient would be counted in the SLEDAI count.

Similarly, the proportion of responders to SLEDAI-4 at treatment completion will be analyzed using logistic regression model as specified for the primary analysis in Section 4.4.1.

# 4.6. Supplementary Estimands for Primary and Secondary Objectives

A supportive estimand for the primary and secondary objectives will be considered to address a clinical question: What is the difference between LY3361237 and placebo in the target patient population, in achieving successful response at Week 24 without regards to violation of concomitant medication rules?

The primary and secondary objective will be additionally assessed, under a situation when the use of concomitant medications may violate the specified rules, but best effort is made to

comply, through a supplementary estimand. Multiple ICE strategies will be applied to construct this supplementary estimand. The ICE – "intervention discontinuation for any reason" – will be handled through the endpoint definition using the composite variable strategy, and all other ICEs including "any concomitant medication violation" will be handled using the treatment policy strategy. The supplementary estimand for primary objective is described by the following attributes:

**Population:** participants with moderate to severe SLE who present with arthritis and/or rash at baseline. Further details can be found in Protocol BT01 Section 5.

**Endpoint:** responder at Week 24 defined as achieving both of the following criteria:

- achieves remission of arthritis and/or rash at Week 24 as measured by SLEDAI-2K and defined in Protocol BT01 Section 8.1.1, and
- does not permanently discontinue study intervention for any reason prior to Week 24.

**Treatment condition:** study intervention as randomized with best effort to manage use of concomitant medication. Further details on study interventions and concomitant medications can be found in Protocol BT01 Section 6.

**Population-level summary:** unconditional difference in proportions of responders at Week 24 between treatment conditions (LY3361237 vs. placebo).

The analytical approach followed will be similar to Section 4.4.1 after taking into account the ICE strategy described above. The secondary estimands described in Section 4.5 may also be considered for analysis using the aforementioned estimand strategy.

### 4.7. Exploratory Estimands



### 4.7.1. Rash and Arthritis

The change of rash status in patients, as defined by the SLEDAI-2K, at Week 24 will be listed. Specifically, the number of patients with improvement of rash, no change in rash, and worsening of rash will be reported respectively. A Cochran-Mantel-Haenszel test will be used to test between the status of rash (improvement, no change, or worsening) and the treatment group (LY or placebo), with stratification factors based on

- CCI
- CCI

· CCI

For sensitivity analysis, Fisher's exact test will be used to test between the status of arthritis (improvement, no change, or worsening) and the treatment group (LY or placebo).

The change of arthritis status in patients, as defined by the SLEDAI-2K, at Week 24 will be listed. Specifically, the number of patients with improvement of arthritis, no change of arthritis, and worsening of arthritis will be reported respectively. A Cochran-Mantel-Haenszel test will be used to test between the status of arthritis (improvement, no change, or worsening) and the treatment group (LY or placebo), with stratification factors based on:

- CCI
- CCI
- CCI

For sensitivity analysis, Fisher's exact test will be used to test between the status of arthritis (improvement, no change, or worsening) and the treatment group (LY or placebo).

# 4.7.2. Rash and/or Arthritis with Intercurrent Events Handled Using Treatment Policy Strategy

The analysis for the proportion of patients with rash and/or arthritis at Week 24 with the stratification at randomization variables, will be performed as described in the section above for mITT patient population with the ICEs handled using treatment policy strategy as described in Section 4.6. That is, all mITT patients will be analyzed without considering rescue medication use, corticosteroid tapering requirement, or any other possible ICEs.

### 4.7.3. Corticosteroid-Sparing Effect

The proportion of patients receiving ≥10 mg/day prednisone at baseline able to reduce prednisone (or equivalent) dose to ≤7.5 mg for 12 consecutive weeks between Week 12 and Week 24 will be compared between LY3361237 treatment group and placebo. The number and percentage of responders and non-responders at each visit will be presented by treatment group. The number of responders and non-responders will be compared using a chi-square test with respect to the treatment group (LY or placebo). If the number of patients in 1 categorical group in 1 treatment group is less than 5, a Fisher's exact test will be used instead.

# 4.7.4. Individual Organ System Systemic Lupus Erythematosus Disease Manifestations Using Systemic Lupus Erythematosus Disease Activity Index 2000 Components, Cutaneous Lupus Erythematosus Disease Area and Severity Index, and Joint Counts

For SLEDAI-2K, within each organ system and each individual item (as detailed in Section 6.3), the proportion of patients who go from "present" at baseline to "absent" at Week 12 and Week 24 will be compared between treatment group and placebo with a Fisher's exact test. No statistical comparison will be performed for the summaries by individual items.

The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) consists of the disease activity and damage scores. Activity is scored on the basis of erythema, scale/hyperkeratosis, mucous membrane involvement, acute hair loss, and nonscarring alopecia.

Damage is scored in terms of dyspigmentation and scarring, including scarring alopecia. The scores are calculated by simple addition based on the extent of the symptoms. Note that when calculating the total damage score, the dyspigmentation score is multiplied by 2 if dyspigmentation usually lasts >12 months. Both disease activity and damage scores will be summarized by treatment and visit separately.

CLASI change from baseline in the activity and damage scores will be summarized and analyzed at Week 4 through Week 24 by linear regression method as described in Section 4.1. In addition, the change from baseline in proportion of patients with  $\geq$ 50% reduction in the disease activity score and damage scores at Week 12 and Week 24 will be analyzed by a logistic regression model, as described in Section 4.1. This analysis (proportion of patients with  $\geq$ 50% reduction) will be repeated for those patients who had a baseline CLASI activity score of 10 or higher.

The number of tender and swollen joints will be determined by examination of 28 joints (14 joints on each side of the patient's body). These 28 joints will be assessed and classified as no symptoms, tender only, swollen only, tender and swollen, or not evaluable. The number of tender and swollen joints ranges from 0 to 28, respectively.

Joints will be assessed for tenderness by pressure and joint manipulation on physical examination. Any positive response on pressure, movement, or both will then be translated into a single tender versus nontender dichotomy. Joints will be classified as either swollen or not swollen. Swelling is defined as palpable fluctuating synovitis of the joint. Swelling secondary to osteoarthrosis will be assessed as not swollen, unless there is unmistakable fluctuation. The change from baseline in the number of 28 tender and swollen joint counts affected by SLE arthritis at Week 4 through Week 24 will be summarized and analyzed by linear regression as described in Section 4.1. The proportion of patients with  $\geq$ 50% reduction in the number of tender/swollen joints affected by SLE arthritis at Week 12 and Week 24 will also be performed by logistic regression as described in Section 4.1. This analysis (proportion of patients with  $\geq$ 50% reduction) will be repeated for those patients who had a baseline count of tender joints  $\geq$ 8 and a baseline count of swollen joints  $\geq$ 8.

Imputation rules for SLEDAI-2K and joint count are described in Sections 6.3 and 6.5, respectively.

### 4.7.5. Lupus Low Disease Activity State

A lupus low disease activity state (LLDAS) response is defined as a low level of disease activity attained with or without use of low-dose steroids and/or tolerated standard maintenance doses of standard of care immunosuppressant medications<sup>4</sup>. In detail, the definition of LLDAS is

- 1. SLEDAI-2K ≤4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity
- 2. no new lupus disease activity compared with the previous assessment
- 3. a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI PGA (scale 0-3) ≤1
- 4. a current prednisolone (or equivalent) dose ≤7.5 mg daily, and

well-tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.

The proportion of patients who achieve LLDAS at Week 24 will be compared between LY3361237 treatment group and placebo. The number and percentage of responders and non-responders at each visit will be presented by treatment group. The proportion of responders will be compared using a logistic regression model as specified in Section 4.1.

### 4.7.6. British Isles Lupus Assessment Group-Based Composite Lupus Assessment

The proportion of patients who meet criteria for response as defined by BILAG-based Composite Lupus Assessment (BICLA) at Week 24 will be compared between LY3361237 treatment group and placebo. The eligibility criteria for BICLA assessment for the mITT patients are:

- BILAG 2004 index level A disease activity in ≥1 organ system at baseline, or
- BILAG 2004 index level B disease activity in ≥2 organs systems if no level A disease activity was present at baseline.

The BICLA is a composite index used to assess disease activity in SLE. A BICLA response is defined as follows:

- reduction of all baseline BILAG-2004 A to B or C or D; and baseline BILAG-2004 B to C or D; and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B
- no worsening from baseline in SLEDAI-2K, where worsening is defined as any increase from baseline in SLEDAI-2K, and
- no worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.3 points on PGA of Disease Activity.

The number and percentage of responders and non-responders at each visit will be presented by treatment group. The proportion of responders will be compared using a logistic regression model as specified in Section 4.1.

### 4.7.7. Physician's Global Assessment of Disease Activity

PGA scores will be summarized by treatment group and visit using descriptive statistics (n, mean, SD, median, minimum, and maximum). Similarly, the change from baseline in PGA scores will be summarized at all scheduled postbaseline visits. The change from baseline score to each scheduled visit will be analyzed using an linear regression model as described in Section 4.1.

### 4.7.8. Time to, and Incidence of, Any Flare and First Severe Flare

| Cox regression model will be used for the time-to-event analyses. |
|---|
| The Kaplan-Meier estimate of the proportion of |
| patients experiencing severe/mild/moderate flare will be presented for each severity. The |
| Kaplan-Meier estimate of the proportion of patients experiencing flare regardless of the severity |

will also be presented. Estimates and 90% CIs for the 25th percentile, median, and 75th percentile will be provided, if estimable, by treatment group.

### 4.7.9. Serologic Markers of Systemic Lupus Erythematosus

In patients with elevated anti-double stranded DNA (anti-dsDNA) at baseline, proportion of patients with normal/high at Week 12 and Week 24 will be analyzed using Fisher's exact test.

In patients with elevated anti-dsDNA at baseline, change in anti-dsDNA level at Week 4 through Week 24 compared to baseline will be analyzed using linear regression model as described in Section 4.1.

In patients with low complement 3 (C3) at baseline, proportion of those who become normal/high at endpoint (Week 12 and Week 24) will be analyzed using Fisher's exact test.

In patients with low complement 4 (C4) at baseline, proportion of those who become normal/high at endpoint (Week 12 and Week 24) will be analyzed using Fisher's exact test.

In patients with low C3 and C4 at baseline, change in C3 and C4 levels at Week 4 through Week 24 compared to baseline will be analyzed using linear regression model as described in Section 4.1.

### 4.7.10. Interferon Gene Signature

Interferon Signature Genes (ISGs) are a large set of genes that are induced in target cells by type 1 interferons.

# 4.7.11. Systemic Lupus Erythematosus International Collaborating Clinics Damage Index

The change from baseline to Week 24 will be analyzed using linear regression with LOCF as the imputation method as described in Section 4.1. Details of the Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) Damage Index score are provided in Section 6.6.

### 4.8. Safety Analyses

See Master Study IMMA SAP (Section 4.10) for safety assessments and safety monitoring activities required for all ISAs. Procedures specified in the following subsections of this ISA must be followed in addition to those described in Master Protocol IMMA.

All safety data will be descriptively summarized by treatment groups (LY and placebo) and analyzed based on the safety population described in Section 3. The safety analyses include AEs, safety in special groups and circumstances, laboratory analytes, the 16-Item Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR16), the Columbia Suicide Severity Rating Scale (C-SSRS), electrocardiograms, and vital signs. The duration of exposure will also be summarized. The categorical safety measures will be summarized using descriptive measures and may be analyzed by Fisher's exact test. The mean change in the continuous safety measures

including vital signs, QIDS-SR16, physical characteristics, and laboratory values will be summarized by visits and analyzed by linear regression, with treatment and baseline values in the model. More details are provided in subsequent sections.

For infections, an IR per 100 patient-years of observation (PYO), will be provided. PYO will be calculated as the sum of all patient observation time in the treatment group. For a patient with an event, the observation time will end at the first event date; for a patient without the event, the observation time will be censored at the patient's last treatment dose date plus 30 days or the patient's last visit, whichever occurs first. Only events that occur within 30 days after the patient's treatment discontinuation date will be considered.

See formula as follows:

$$PYO = \sum_{pt \ w \ event} \frac{event \ start \ date - first \ trt \ dose \ date + 1}{365.25} \\ + \sum_{pt \ w/o \ event} \frac{last \ observation \ date - first \ trt \ dose \ date + 1}{365.25}$$

IR will be calculated as follows:

$$IR = \frac{unique\ number\ of\ patients\ with\ at\ least\ an\ event}{PYO} x100$$

For each IR provided, a 95% CI will be calculated based on the Poisson distribution. Treatment group comparisons (LY and placebo) based on IR will be provided based on the incidence rate difference together with its 95% CI.

Not all displays described in this section will necessarily be included in the CSRs. Any display described and not provided in the CSR would be available upon request. Not all displays will necessarily be created as a "static" display. Some may be incorporated into interactive display tools instead of or in addition to a static display. Any display created interactively will be included in the CSR if deemed relevant to the discussion.

### 4.8.1. Extent of Exposure

Duration of exposure to study drug will be summarized for the safety population by treatment group. Exposure will be calculated as the date of last dose of study drug (or date of discontinuation) minus the date of first dose of study drug plus 1 day. Total patient-years (PYs) of exposure will be reported for each treatment group for overall duration of exposure. Descriptive statistics (n, mean, SD, minimum, first quartile, median, third quartile, and maximum) will be provided for patient-days of exposure and the frequency of patients falling into different exposure ranges will be summarized. Exposure ranges are as follows:

- ≥4 weeks, ≥12 weeks, and ≥24 weeks, and
- >0 to <4 weeks, >4 weeks to <12 weeks, >12 weeks to <24 weeks, and >24 weeks.

Overall exposure will be summarized in total PYs, which are calculated according to the following:

Exposure in PYs = sum of duration of exposure in days (for all patients in treatment group) / 365.25

No p-values will be reported in these tables as they are intended to describe the characteristics of the study sets.

### 4.8.2. Adverse Events

### 4.8.2.1. Adverse Events

AEs are recorded in the eCRF. Each AE will be coded to SOC and PT, using the MedDRA version that is current at the time of database lock. Severity of AEs is recorded as mild, moderate, or severe.

Treatment-emergent adverse events (TEAEs) are defined as events that either first occurred or worsened in severity after the first dose of study drug and the earliest of the visit study drug disposition date or the last visit date during the treatment period, whichever occurred first, and up to 30 days after study treatment discontinuation. The MedDRA Lowest Level Term (LLT) will be used in defining which events are treatment-emergent. The maximum severity for each LLT during the baseline period until the first dose of the study medication will be used as baseline. If an event is preexisting during the baseline period, but it has missing severity, and the event persists during the treatment period or up to 30 days after treatment discontinuation, then the baseline severity will be considered mild for determining any postbaseline treatmentemergence (that is, the event is treatment-emergent unless the severity is coded mild at postbaseline). If an event occurring postbaseline has a missing severity rating, then the event is considered treatment-emergent. Should there be insufficient data for an AE start date to make this comparison (for example, the AE start year is the same as the treatment start year, but the AE start month and day are missing), the AE will be considered treatment-emergent. For events occurring on the day of the first dose of study treatment, the day and time of the onset of the event will both be used to distinguish between pretreatment and posttreatment in order to derive treatment-emergence.

In general, summaries will include the number of patients in the safety population (N), frequency of patients experiencing the event (n), and relative frequency (that is, percentage; n/N\*100).

In an AE overview table, the number and percentage of patients in the safety analysis set who experienced death, a serious adverse event (SAE), any TEAE, permanent discontinuation from study drug due to an AE, temporary interruption of study drug due to an AE or laboratory abnormality, or a severe TEAE will be summarized by treatment group.

The number and percentage of patients with TEAEs will be summarized by treatment group in the 2 formats listed below:

 by MedDRA PT nested within SOC with SOCs ordered alphabetically, and events ordered within each SOC by decreasing frequency in the LY3361237 450 mg treatment group, and  by MedDRA PT with events ordered by decreasing frequency in the LY3361237 450 mg treatment group.

For events that are gender specific, the denominator and computation of the percentage will only include patients from the given gender.

AEs leading to permanent discontinuation of study drug and AEs leading to temporary interruption of study drug will also be summarized by treatment group using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3361237 450 mg treatment group.

A summary of temporary interruptions of study drug will also be provided, showing the number of patients who experienced at least 1 temporary interruption and the number of temporary interruptions per patient with an interruption. Furthermore, the duration of each temporary interruption (in days) and the cumulative duration of dose interruption (in days) using basic descriptive statistics (n, mean, SD, minimum, first quartile, median, third quartile, and maximum) will be displayed.

Common TEAEs are defined as TEAEs that occurred in ≥2% (before rounding) of patients in any treatment group including placebo. The number and percentage of patients with common TEAEs will be summarized by treatment using MedDRA PT ordered by decreasing frequency in the LY3361237 450 mg treatment group.

The number and percentage of patients with TEAEs will be summarized by maximum severity by treatment using MedDRA PT ordered by decreasing frequency for the common TEAEs and by treatment group using MedDRA PT nested within SOC, respectively. Events will be ordered by decreasing frequency within SOC in the LY3361237 450 mg treatment group. For each patient and TEAE, the maximum severity for the MedDRA level being displayed is the maximum postbaseline severity observed from all associated LLTs mapping to that MedDRA PT.

### 4.8.2.2. Serious Adverse Events

An individual listing of all SAEs including preexisting conditions will be provided. A separate listing will include AEs that led to permanent discontinuation from the study drug. In addition, a listing of AEs that occur more than 30 days after study treatment discontinuation will be provided.

With the ICH E2A guideline, an SAE is any AE that results in 1 of the following outcomes:

- death
- initial or prolonged inpatient hospitalization
- a life-threating experience (that is, immediate risk of dying)
- persistent or significant disability/incapacity
- congenital anomaly/birth defect, or
- considered significant by the investigator for any other reason.

The number and percentage of patients who experienced any ICH-defined SAE will be summarized by treatment group during the treatment and follow-up periods using MedDRA PT nested within SOC. Events will be ordered by decreasing frequency within SOC in the LY3361237 450 mg treatment group. In addition, the SAEs will be summarized by treatment group using MedDRA PT without SOC. An individual listing of all SAEs will be provided.

### 4.8.3. Adverse Events of Special Interest

### 4.8.3.1. Infections

Completion of the Infection eCRF page is required for each infection reported as an AE or SAE.

Infections will be defined using all PTs from the MedDRA Infections and Infestations SOC. Serious infection will be defined as all the infections that meet the SAE criteria.

The number and percentage of patients with TEAEs of infections, serious infections, and infections resulting in study drug discontinuation will be summarized by treatment group using McdDRA PTs.

The number and percentage of patients with TEAEs of infections by maximum severity will be summarized by treatment group using MedDRA PTs.

For infections of special interest (herpes zoster, and herpes simplex), serious infections, and potential opportunistic infections (POIs) the IR and 95% CI will be calculated (for detail, see Section 4.8).

Treatment-emergent infectious events will be reviewed in context of other clinical and laboratory parameters. A listing of patients experiencing treatment-emergent infectious AEs will be provided. The listing will include patient demographics, treatment group, treatment start and stop dates, infectious event, event start and stop dates, total leukocytes, total lymphocytes, absolute neutrophils, event seriousness, and event outcome.

The infectious TEAE will be further analyzed in terms of potential opportunistic infection, herpes zoster, and herpes simplex. A summary of hepatitis B virus (HBV) DNA monitoring results and association between infection and neutropenia/lymphopenia will also be provided in the context of infections.

### Potential opportunistic infections

The sponsor will identify infections considered to be opportunistic based on the article by Winthrop et al. (2015). See also Master Protocol IMMA (Appendix 10.5).

POIs will be identified in 2 ways3:

- 1. POIs will be identified from TEAEs based on a Lilly-defined list of MedDRA PTs shown in Section 6.9. The list is maintained outside Study BT01 SAP and can be updated without an amendment to Study BT01 SAP. These PTs are a subset of terms from the Infections and Infestations SOC.
- Medical will review the list of POIs, including the details captured on the infectionspecific eCRF, and determine whether the infection is a 'confirmed opportunistic infection'.

The summary analysis of opportunistic infections identified using the 2 approaches above will be provided. Events will be ordered by decreasing frequency of pathogen nested under pathogen species (mycobacteria, bacteria, fungal, viral, and parasites). The order of frequency will be determined using the LY3361237 450 mg group.

### Herpes zoster

A summary table of herpes zoster will be provided. Herpes zoster will be defined based on the MedDRA PTs as listed under Herpes zoster (any form) (II) in Section 6.9, excluding Varicella virus test (10070444). The summary table will also include event maximum severity, seriousness, whether resulting in temporary study drug interruption, whether resulting in study drug discontinuation, whether treated with antiviral medication, and event outcome.

If a patient has more than 1 event of herpes zoster, the event with the maximum severity will be used in these summary tables. If more than 1 event of herpes zoster occurs with the same severity, the event with the longest duration will be used in the summary table.

### Herpes simplex

A summary analysis of herpes simplex will be provided. Herpes simplex will be defined based on the MedDRA PTs as listed under Herpes simplex (invasive disease only) (IV) in Section 6.9. The summary table will include event maximum severity, seriousness, whether resulting in temporary study drug interruption, whether resulting in study drug discontinuation, and whether treated with antiviral medication. Antiviral medication will be selected based on Anatomical Therapeutic Chemical code level 2 "antiviral for systemic use."

If a patient has more than 1 event of herpes simplex, the event with the maximum severity will be used in these summary tables. If more than 1 event of herpes simplex occurs with the same severity, the event with the longest duration will be used in the summary table.

### Hepatitis B virus DNA

A listing of patients with detectable HBV DNA will be provided.

HBV DNA status (not detectable, detectable but not quantifiable [that is, <29 IU/mL], and quantifiable [that is, ≥29 IU/mL]) will be summarized by treatment group stratified by baseline HBV serology status, specifically:

- HBsAb-/HBcAb-
- HBsAb+ / HBcAb-
- HBsAb+ / HBcAb+, and
- HBsAb-/HBcAb+.

### Association between infection and neutropenia/lymphopenia

To evaluate the association between infection and neutropenia and/or lymphopenia, the frequency of infections will be provided by the worst Common Terminology Criteria for Adverse Events (CTCAE) grades of neutropenia and lymphopenia, respectively. Infection outcomes considered for this analysis are any treatment-emergent infection, serious infection, and herpes zoster. For this analysis, no statistical comparison will be provided.

In addition, a summary table will be provided for treatment-emergent infections that were preceded or accompanied by neutropenia/lymphopenia. For this analysis, neutropenia is defined as CTCAE Grade 2 or greater. Infection events with onset date ≤14 days before or after the Grade 2 neutrophil/lymphocyte count collection date will be considered as infections preceded or accompanied by neutropenia.

### 4.8.3.2. Systemic Hypersensitivity Reactions

Many drugs, but particularly biologic agents, carry the risk of systemic hypersensitivity reactions. If such a reaction occurs, additional data describing each symptom should be provided to the sponsor in the eCRF.

Sites should have appropriately trained medical staff and appropriate medical equipment available when the study participants are receiving the study intervention. It is recommended that participants who experience a systemic hypersensitivity reaction be treated per national and international guidelines.

### Sample collection at time of systemic hypersensitivity events

In the case of generalized urticaria or anaphylaxis, additional samples should be collected as described in Protocol BT01 Attachment 10.1.2. Laboratory results are provided to the sponsor via the central laboratory.

There are two time periods:

- time period A, potential immediate hypersensitivity: analysis of TEAEs occurring on the day of study drug administration, and
- time period B, potential non-immediate hypersensitivity: analysis of TEAEs occurring strictly after the day of study drug administration (but prior to subsequent drug administration).

Analyses of both time periods use current Standardised MEDdra Queries (SMQs), published by the Maintenance and Support Services Organization, to search for relevant events. The TEAEs are characterized as follows:

- Anaphylactic reaction SMQ (20000021; narrow, algorithm per SMQ guide, and broad)
- Hypersensitivity SMQ (20000214; narrow and broad), and
- Angioedema SMQ (20000024; narrow and broad).

Identified events will be listed, by temporal order within patient ID, and will include SOC, PT, SMQ event categorization including detail on the scope (narrow or broad), reported AE term, AE onset and end dates, severity, seriousness, outcome, and so on.

### 4.8.4. Injection Site Reaction

The number and percentage of patients who experienced injection site reactions (ISR) will be summarized by treatment group and by visit. The number and percentage of patients with the following ISR records will be summarized by treatment group and by visit:

anatomical location of the ISR

- abdomen side
- directionality of the anatomical location of the administration
- arm side
- thigh side
- whether the subject has any injection site erythema (reddening)
- severity of the injection site erythema
- whether the subject has any injection site induration (hardening or thickening of tissue)
- severity of the injection site induration
- whether the subject has any injection site pain (including burning)
- severity of the injection site pain
- whether the subject has any injection site pruritus
- severity of the injection site pruritus
- whether the subject has any injection site edema (swelling or accumulation of fluid in tissues at height above normal skin)
- severity of the injection site edema, and
- injection related event occur, in relationship to the study treatment (time to onsite of ISR)

If an ISR is reported by a participant or site staff, the ISR CRF will be used to capture additional information about this reaction (for example, injection-site pain, degree and area of erythema, induration, pruritis, and edema).

### 4.8.5. Clinical Laboratory Evaluations

Please refer to Section 4.10.4 in Study IMMA SAP.

### 4.8.6. Vital Signs and Other Physical Findings

Please refer to Section 4.10.5 in Study IMMA SAP.

### 4.8.7. Depression and Suicide

Please refer to Section 4.10.6 in Study IMMA SAP.

### 4.9. Other Analyses

### 4.9.1. Concomitant Therapy

Previous and concomitant medications will be summarized by treatment for each ISA and will be presented by Anatomical Therapeutic Chemical drug classes using the WHO Drug Dictionary version WHODDMAR19B3 (Uppsala Monitoring Centre 2019). Details can be found in Master Protocol IMMA Section 6.5 and Protocol BT01 Section 6.5. When the primary estimand is used for analyses, participants who require initiation or increase in dosage of corticosteroids, antimalarials, or immunosuppressants after randomization will be analyzed as non-responders from the day of initiation or increase in medication.

This describes how, for the efficacy analyses with primary estimand, the participant's responder/non-responder status will be handled in cases of such medication changes.

| If the following medication is started after baseline or is increased in dosage after baseline | Then the participant's status for the efficacy analyses, from the time of change onward, will be: |
|---|---|
| Corticosteroid | Non-responder |
| Antimalarial | Non-responder |
| Immunosuppressant (from the list in the protocol) | Non-responder |

### 4.9.2. Treatment Compliance

Treatment compliance with study intervention will be summarized by treatment group. A participant will be considered significantly noncompliant if he or she fails to receive the study intervention within the required treatment window as defined in Protocol BT01 Section 1.3, Figure 1. Overall compliance with therapy is defined to be missing no more than 20% of the expected injections and not missing 2 consecutive dosing visits.

Treatment compliance with study medication will be assessed from the randomization visit (Week 0) to Visit 14 (Week 24) during the treatment period. Compliance will be summarized from randomization until end of treatment using the mITT population. Compliance to study drug in the period of interest will be calculated as follows:

$$\frac{\text{actual total # of injections}}{\text{Expected total # of injections}} * 100.$$

The summary statistics of the percent of compliance and noncompliance rate will be summarized by treatment group. The percent of compliance for Week 0 (Visit 2) through Week 24 (Visit 14) will be presented, along with the associated noncompliance rates.

### 4.9.3. Immunogenicity Assessments

The frequency and percentage of participants with preexisting ADAs and with treatmentemergent ADAs (TE ADAs) to LY3361237 will be tabulated and listed.

For participants who are ADA negative at baseline, TE ADAs are defined as those with a titer 2-fold (1 dilution) greater than the minimum required dilution (1:10) of the assay (treatment-induced ADAs). For participants who are ADA positive at baseline, TE ADAs are defined as

those with a 4-fold (2 dilution) increase in titer compared to baseline (treatment-boosted ADAs). For the TE ADA positive participants, the distribution of maximum titers will be described.

The relationship between the presence of antibodies to LY3361237 and the LY3361237 serum concentrations and receptor occupancy (RO) response, including safety and efficacy of LY3361237, may be assessed to show participants with ADA titers versus those without titers.

### 4.9.4. Patient-Reported Outcomes

For analysis of QIDS-SR16 data, see the methods described for safety data in Section 9.3.5 of the Master Protocol IMMA. If additional PROs are considered, dichotomous variables will be analyzed using logistic regression analyses, whereas linear regression will be the primary method of analysis for continuous endpoints. The analyses will be based on the mITT population, unless otherwise specified.

### 4.9.5. Subgroup Analyses

Subgroup analyses may be conducted for the primary endpoint rash and/or arthritis remission at Week 24 using the mITT population. Subgroups that may be evaluated include interferon gene signature status, original genetic sex, race, geographic region, baseline anti-dsDNA status, baseline SLEDAI-2K, complement status, previous therapies, and disease duration.

In detail, the following subgroups (but not limited to only these) may be evaluated:

- gender (male; female)
- baseline anti-dsDNA status (positive; negative)
- baseline interferon signature (positive; negative)
- baseline complement (low C3 and/or low C4; normal/high C3; normal/high C4)
- race (Asian; Black/African American; White; other)
- disease severity at baseline (SLEDAI-2K): (<10; ≥10)</li>
- region (United States; Europe; rest of the world), and
- corticosteroid dose at baseline: (<10 mg; ≥10 mg).</li>

If the number of participants is too small (less than 5 participants) within a subgroup, then the subgroup categories may be redefined prior to unblinding the study. Descriptive statistics will be provided for each treatment and stratum of a subgroup. Categorical variables will be analyzed individually with a logistic model that contains the treatment, the subgroup variable, and subgroup by treatment interaction. The treatment-by-subgroup interaction will be tested at the 10% significance level to determine whether treatment differences are the same for each subgroup category. For the continuous variables, if the subgroup analyses are conducted only at Week 24 (Visit 14), linear regression model with LOCF will be used, in which the treatment, the baseline values, the subgroup variable, and subgroup by treatment interaction will be included as covariates in the model. For the categorical variables, the number of responders and response rate may be reported for each subgroup.



Additional analyses may be performed as deemed necessary. If applicable, any early access will be detailed in the Unblinding Plan.

### 4.10.1. Assessment Committee

If an interim analysis is conducted, it will be performed by an internal assessment committee (AC). Details of the planned interim data analyses and the AC data review process are included in the Study BT01 AC charter.

### 4.11. Pharmacokinetic Assessment



# 4.13. Data Monitoring Committee

Not applicable. An internal AC will be used to conduct the interim analysis.

Details of the planned interim data analyses and the AC data review process are included in an AC charter.

# 4.14. Changes to Protocol-Planned Analyses

There were no changes from the protocol specified statistical analysis.
# 5. Sample Size Determination

In this ISA, approximately 180 patients will be screened to achieve 90 participants randomly assigned to study intervention (45 per treatment group).

The sample size calculation is based on the primary efficacy endpoint, remission of rash and/or arthritis as assessed by SLEDAI-2K at Week 24. Approximately 90 participants will be randomized in a 1:1 ratio to LY3361237 450 mg and placebo treatment groups.

# 6. Supporting Documentation

# 6.1. Appendix 1: Description and Derivation of Efficacy Outcomes Measures and Endpoints

Table APP.1.1. Description and Derivation of Efficacy Outcomes Measures and Endpoints

| Measure | Description | Variable | Derivation/Comment | Definition of Missing |
|---|---|---|---|---|
| SLEDAI-<br>2K | The SLEDAI-2K is a global disease activity instrument that focuses on high-impact disease manifestations across 9 organ domains: constitutional, mucocutaneous, musculoskeletal, vascular, cardiorespiratory, CNS, immunologic, renal, and hematologic. | SLEDAI-<br>2K Total<br>Score | Calculated by summing the weighted organ manifestation. | Any item scores are missing (not done, not assessed, NA or empty), but the visit occurred. Baseline data for that item can be carried forward from the last nonmissing data during the screening period. Postbaseline data for that item can be carried forward from the last nonmissing data if that data is obtained within the previous 34 days of that visit. After imputation, If any item is still missing at the baseline visit, it will be imputed as 0. For Renal domain, if urinary casts, hematuria and pyuria items are still missing for any postbaseline visit, they will be |
| | | Individual Organ Domain Improveme nt Defined by SLEDAI- 2K Individual Organ Domain No Worsening | Patients with SLEDAI-2K score >0 within the organ domain at baseline, and able to decrease SLEDAI-2K (from baseline) within each organ domain score, separately. Among patients with at least one SLEDAI-2K item = 0 (not present) in the organ domain score at | imputed as 0. Missing if any SLEDAI-2K item for that organ domain remains missing after instrument level imputation rules are applied. Missing if any SLEDAI-2K item for that organ domain remains missing after |

| | | Defined by<br>SLEDAI-<br>2K<br>No<br>worsening<br>from | baseline, no increment of SLEDAI-2K organ domain score from baseline within each organ domain score, separately. No increment from baseline of >0 points in SLEDAI-2K | instrument level imputation rules are applied. Missing if any SLEDAI-2K item for that organ domain remains missing after |
|---|---|---|---|---|
| | | baseline in<br>SLEDAI-<br>2K | | instrument level imputation rules are applied. |
| SLEDAI-4 | SLEDAI-4 is an index to measure overall improvement in disease activity (SLEDAI-2K) | SLEDAI-4<br>Responder | A ≥4-point reduction in SLEDAI-2K score from baseline. | Missing if SLEDAI-2K<br>total score is missing after<br>instrument level imputation<br>rules are applied. |
| SRI-4 | SRI-4 is a composite index to measure overall improvement in disease activity (SLEDAI-2K) while ensuring there is no worsening in other organ systems (BILAG and PGA) | SLE<br>Responder<br>Index 4 | <ul> <li>A decrease in SLEDAI-2K ≥4 (from baseline)</li> <li>No new BILAG A and no more than 1 new BILAG B disease activity score / organ domain (both compared with baseline), and</li> <li>No worsening in PGA (defined as an increase of 0.3 points [10 mm] from baseline)</li> </ul> | After each instrument level imputation rule is applied and there is still at least one missing component, if the nonmissing components are all 'Y' then SRI-4 is missing. if any of the nonmissing component is 'N' then the SRI-4 is 'N.' |
| BILAG-<br>2004 | BILAG-2004 assesses 97 clinical signs, symptoms and laboratory parameters across 9 organ system domains: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and hematological | BILAG | A, B, C, D, or E score will be used in analyses for each of the 9 individual organ systems. | Within each organ domain (except renal and hematological), any missing data will be assumed to be 'Not present' if there is at least 1 nonmissing item in that organ. If all items in one organ domain are completely missing but the visit occurred, then the letter score of that organ from the previous visit will be pulled forward, provided data were obtained within 34 days of visit; otherwise missing except when the letter score from the last nonmissing visit is E, then E score will be pulled forward. |

| BIL | AG ovemen Reduction of all baseline BILAG B/C/D and basel BILAG B to C/I No BILAG wors in other organ sy where worsening defined as ≥1 ne BILAG A or ≥2 BILAG B | missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the missing is at the baseline (any one or all |
|---|---|---|
|---|---|---|

| | | No BILAG worsening Individual Organ Domain Improveme nt Defined by BILAG | No new BILAG A and no more than 1 new BILAG B disease activity score (both compared with baseline), where worsening is defined as ≥1 new BILAG A or ≥2 new BILAG B, both compared with the baseline. The baseline BILAG A improved to BILAG B at the visit will not be considered as the new BILAG B. Among patients with BILAG A or B at baseline and able to reduce the baseline BILAG A to B/C/D and BILAG B to C/D for each organ domain, separately. | For the no worsening part, missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the baseline (any one or all domains) is BILAG A and the value at the visit is missing, then the other nonmissing organ domains will be used to determine the response status. If both components are missing or one component is missing and the other one is 'Y,' then missing. If at least one component is 'N', then 'N.' Missing if any of 9 domains at baseline or at the visit remains missing after instrument level imputation rules are applied except when the baseline (any one or all domains) is BILAG A and the value at the visit is missing, then the other nonmissing organ domains will be used to determine the response status. Missing if baseline or value remains missing after instrument level imputation rules are applied. |
|---|---|---|---|---|
| | | Individual<br>Organ<br>Domain No<br>Worsening<br>Defined by<br>BILAG | separately. Among patients without BILAG A at baseline, no increment of baseline BILAG B/C/D/E to A and baseline BILAG C/D/E to B for each organ domain, separately. | Missing if baseline or value remains missing after instrument level imputation rules are applied. |
| PGA | The PGA is the physician's assessment of the | PGA score<br>PGA<br>category | Permitted range of values is from 0 to 100 mm. | If the visit occurred, data can be carried forward if |

| | patient's overall disease activity due to SLE. It is scored using a visual analog scale where 0 mm indicates no disease activity and 100 mm indicates the most severe disease activity possible. There are benchmarks of 0 (0 mm), 1 (33 mm), 2 (67 mm), and 3 (100 mm) on the line | No<br>worsening<br>in PGA | PGA categories are defined as: None (0) = '0 mm', Mild (>0 and <1.5) = '>0 to <50 mm', Moderate (≥1.5 to ≤2.5) = '≥ 50 mm to ≤83 mm', Severe (>2.5) = '>83 mm'. Worsening is defined as an increase of ≥0.3 points (10 mm) from baseline. Therefore, no worsening is defined as any decrease, no change, or <0.3 points (10 mm) increase from baseline. | obtained within 34 days of visit; otherwise missing. Missing if baseline or value remains missing after instrument level imputation rules are applied. |
|---|---|---|---|---|
| | corresponding to no,<br>mild, moderate, and<br>severe SLE disease<br>activity, respectively. | PGA ≤1 | PGA ≤33 mm | Missing if value remains<br>missing at the visit after<br>instrument level imputation<br>rules are applied. |
| BICLA | BICLA is a composite index to measure overall improvement in disease activity (BILAG) while ensuring there is no worsening in other organ systems (SLEDAI and PGA) | BILAG<br>Based<br>Composite<br>Lupus<br>Assessment | BILAG Improvement Reduction of all baseline BILAG A to B/C/D and baseline BILAG B to C/D No BILAG worsening in other organ systems, where worsening is defined as ≥1 new BILAG A or ≥2 New BILAG B No worsening from baseline in SLEDAI-2K, where worsening is defined as an increase of >0 points from baseline in SLEDAI-2K No worsening from baseline in participants' lupus disease activity, where worsening is defined by an increase ≥0.30 points on a 3-point PGA VAS. | After each instrument level imputation rule is applied and there is at least one component missing, if the nonmissing components are all 'Y' then BICLA will be missing. If any of the nonmissing component is 'N' then the BICLA is 'N.' |
| CLASI | The CLASI is a validated instrument to assess cutaneous | Total<br>Activity<br>Score | Calculated within tablet system with edit checks; no additional derivation. | Within tablet system: If any item scores, but not all are |

| | manifestations of SLE consisting of 2 scores: | Total<br>Damage<br>Score | Calculated within tablet system with edit checks; no additional derivation. | missing then impute a score of 0 for the missing item(s). For completely missing questionnaires, data can be carried forward if obtained within 34 days of visit; otherwise missing. Within tablet system: if any item scores, but not all are missing then impute a score of 0 for the missing item(s). For completely missing questionnaires, data can be carried forward if obtained within 34 days of visit; otherwise missing. |
|---|---|---|---|---|
| LLDAS | The LLDAS is a composite measure designed to identify patients achieving a state of low disease activity. | LLDAS | <ul> <li>SLEDAI-2K ≤ 1, with no activity in SLEDAI-2K major organ systems (CNS, Vascular, Renal, Cardiorespiratory and Constitutional), where "no activity" is defined as all items of SLEDAI-2K within these major organ systems equal to 0.</li> <li>No new features of Lupus disease activity in SLEDAI-2K compared to previous occurred visit, where the "new feature" is defined as any of the SLEDAI-2K 24 items changed from 0 to greater than 0.</li> <li>PGA ≤1</li> <li>Current prednisone or equivalent ≤7.5 mg/day</li> </ul> | After each instrument level imputation rule is applied and there is at least one component missing, if the nonmissing components are all 'Y' then LLDAS will be missing. If any of the nonmissing component is 'N' then the LLDAS is 'N.' |
| SLEDAI<br>Flare Index | The SFI uses the<br>SLEDAI score,<br>disease activity<br>scenarios, treatment<br>changes, and PGA to | SFI Flare | No derivation; used as entered. | The absence of a flare record, or 'Non Applicable,' both are indicative of no occurrence of flare. |
| | define mild/moderate<br>and severe flares. | Time to first<br>flare | Time to first flare will be derived as the first date of most recent flare minus date of first injection plus 1. | Not applicable |

| SLICC/AC | SLICC/ACR Damage | SLICC/AC | Calculated as the sum of all |
|---|---|---|---|
| R | Index assesses | R Damage | available entries with a |
| | damage to 12 organ | Index Score | maximum score of 47. |
| | systems regardless of | | |
| | its cause. | | |

Abbreviations: ACR = American College of Rheumatology; BICLA = British Isles Lupus Assessment Group-based Composite Lupus Assessment; BILAG = British Isles Lupus Assessment Group - 2004; CLASI = Cutaneous Lupus Erythematosus Disease Area and Severity Index; CNS = central nervous system; LLDAS = Lupus Low Disease Activity State; MCS = Mental Component Summary; N = no; NA = not applicable; PCS = Physical Component Summary; PGA = Physician's Global Assessment; PROMIS SF = Patient-Reported Outcomes Measurement Information System Short Form; Q2W = every 2 weeks; SFI = Self-Report Family Instrument; SLE = systemic lupus erythematosus; SLEDAI-2K = Systemic Lupus Erythematosus Disease Activity Index 2000; SLEDAI-4 = a ≥4-point reduction in SLEDAI-2K score from baseline; SLICC = Systemic Lupus Erythematosus International Collaborating Clinics; SRI-4 = Systemic Lupus Erythematosus Responder Index-4; VAS = Visual Analog Scale; Y = yes.

# .2. Appendix 2: Description of Efficacy Analyses

The table below provides the detailed analyses including estimand strategy, analysis method, missing data imputation, analysis population, and analysis type.

Table APP.2.1. Description of Efficacy Analyses

| | | T-11-11 | | | | |
|---|---|---|---|---|---|---|
| Measure | Endpoint | Strategy | Analysis<br>Population | Timepoint | Analysis Method | Analysis Type |
| SLEDAI | SLEDAI-4 | Composite | mITT | LY3471851 vs Placebo | Logistic Regression with | Logistic Regression |
| | | | | at postbaseline visits in | NRI; | with NRI for |
| | | | | the treatment period | Fisher's Exact Test with | Week 24 - Primary |
| | | | | | NRI | Other - Exploratory |
| | | Composite | Per-Protocol | LY3471851 vs Placebo | Logistic Regression with | Exploratory |
| | | | | at postbaseline visits in | NRI; | |
| | | | | the treatment period | Fisher's Exact Test with | |
| | | | | | NRI | |
| | | Treatment | mITT | LY3471851 vs Placebo | Logistic Regression with | Exploratory |
| | | Policy | | at postbaseline visits in | NRI | |
| | | | | the treatment period | Fisher's Exact Test with | |
| | | | | | NRI | |
| | No worsening from | Composite | LLIm | LY3471851 vs Placebo | Logistic Regression with | Exploratory |
| | baseline in | | | at postbaseline visits in | NRI | |
| | SLEDAI-2K | | | the treatment period | Fisher's Exact Test with | |
| | | | | | NRI | |
| | SLEDAI Change<br>from Baseline | Hypothetical | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression | Exploratory |
| | | Composite | mITT | LY3471851 vs Placebo<br>at nostbaseline visits in | linear regression | Exploratory |
| | | | | the treatment period | | |
| | Individual Organ | Composite | mITT - Patients | LY3471851 vs Placebo | Logistic Regression with | Exploratory |
| | Domain | | with SLEDAI-2K | at postbaseline visits in | NRI | |
| | mprovement | | Score / U WILLIAM LINE | uic ucamiciii periou | | |

| | Defined by<br>SLEDAI-2K | | organ domain at<br>baseline | | Fisher's Exact Test with<br>NRI | |
|---|---|---|---|---|---|---|
| | Individual Organ<br>Domain Worsening<br>Defined by<br>SLEDAI-2K | Composite | mITT – Patients with at least one baseline SLEDAI- 2K = 0 in the organ domain at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| | Resolution of Arthritis and/or Rash by SLEDAI- 2K Components | Composite | mITT – Patients with SLEDAI-2K arthritis and/or rash 'Present' at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |
| SRI-4 | SRI-4 | Composite | mITT Per-Protocol | LY3471851 vs Placebo at postbaseline visits in the treatment period LY3471851 vs Placebo at postbaseline visits in the treatment period | Logistic Regression with NRI: Fisher's Exact Test with NRI Logistic Regression with NRI: Fisher's Exact Test with | Logistic Regression<br>with NRJ for<br>Week 24 –<br>Secondary<br>Other – Exploratory<br>Exploratory |
| BICLA | BICLA | Composite | mITT – Patients with at least 1 BILAG A or 2 BILAG B scores at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | NRI<br>Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory |
| | | Composite | Per-Protocol – Patients with at least 1 BILAG A or 2 BILAG B scores at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Exploratory |

| | Ĩ | i i i | j | |
|---|---|---|---|---|
| Logistic Regression<br>with NRI for<br>Week 24 –<br>Secondary<br>Other – Exploratory | Exploratory | Exploratory Exploratory | Exploratory Exploratory | Exploratory |
| Logistic Regression with<br>NRI;<br>Fisher's Exact Test with<br>NRI | Logistic Regression with NRI Fisher's Exact Test with NRI Logistic Regression with NRI | Fisher's Exact Test with NRI Logistic Regression with NRI Fisher's Exact Test with NRI Logistic Regression with NRI Fisher's Exact Test with NRI NRI | linear regression | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI |
| LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo at postbaseline visits in the treatment period LY3471851 vs Placebo at postbaseline visits in | LY3471851 vs Placebo at postbaseline visits in the treatment period LY3471851 vs Placebo at postbaseline visits in the treatment period | LY3471851 vs Placebo at postbaseline visits in the treatment period LY3471851 vs Placebo at postbaseline visits in the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period |
| mITT | mITT – Patients with at least 1 BILAG A or 2 BILAG B at baseline mITT | mITT – Patients with BILAG A or B within the organ domain at baseline mITT – Patients with no BILAG A within the organ domain at baseline | mITT | mITT |
| Composite | Composite<br>Composite | Composite<br>Composite | Hypothetical Composite | Composite |
| LLDAS | BILAG Improvement BILAG No Worsening | Individual Organ Domain - Improvement Defined by BILAG Individual Organ Domain - No Worsening Defined by BILAG | PGA Change from<br>Baseline | No worsening in<br>PGA |
| LLDAS | BILAG | | PGA | |

LY3361237

| | PGA ≤1 | Composite | mITT - Patients | LY3471851 vs Placebo | Logistic Regression with | Exploratory |
|---|---|---|---|---|---|---|
| | | | with PGA > 1 at | at postbaseline visits in | NRI | |
| | | | baseline | the treatment period | Fisher's Exact Test with | |
| CLASI | Total Activity<br>Score, Change<br>from Baseline | Hypothetical | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression | Exploratory |
| | | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression with BOCF | Exploratory |
| | Total Damage<br>Score, Change<br>from Baseline | Hypothetical | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression | Exploratory |
| | | Composite | mITT | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression with BOCF | Exploratory |
| | >50% Reduction in<br>CLASI Total<br>Damage Score | Composite | mITT − Patients with CLASI Total Damage Score ≥10 at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with NRI;<br>Fisher's Exact Test with NRI | Exploratory |
| | ≥50% Reduction in<br>CLASI Total<br>Activity Score | Composite | mITT − Patients with CLASI Total Activity Score ≥10 at baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with<br>NRI | Exploratory |
| Corticoster<br>oid-Sparing<br>Effect | Reduction of prednisone (or equivalent) dose to | Composite | mITT – Patients<br>with prednisone (or<br>equivalent) >10 mg | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Logistic Regression with<br>NRI<br>Fisher's Exact Test with | Exploratory |
| | ≤7.5 mg for 12 consecutive weeks between Week 12 and Week 24 | | at baseline | | NRI | |

| Exploratory | Exploratory | F Exploratory | Exploratory | | F Exploratory | | | | Exploratory | | | | Exploratory | | | Exploratory | | | | Exploratory | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| linear regression | linear regression | linear regression with BOCF | linear regression | | linear regression with BOCF | | | | Logistic Regression with | NRI | Fisher's Exact Test with | NRI | Logistic Regression with | NRI | Fisher's Exact Test with NRI | linear regression | | | | Linear regression with | BOCF | | |
| LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo | the treatment period | LY3471851 vs Placebo | at postbaseline visits in | the treatment period | | LY3471851 vs Placebo | at postbaseline visits in | the treatment period | | LY3471851 vs Placebo | at postbaseline visits in | the treatment period | LY3471851 vs Placebo | at postbaseline visits in | the treatment period | | LY3471851 vs Placebo | at postbaseline visits in | the treatment period | |
| mITT | Per-Protocol | mITT | mITT – Patients<br>with tender ioints | affected by SLE | mITT - Patients | with tender joints | affected by SLE | arthritis at baseline | mITT - Patients | with tender joints | affected by SLE | arthritis at baseline | mITT - Patients | with >8 TJC at | baseline | mITT - Patients | with swollen joints | affected by SLE | arthritis at baseline | mITT - Patients | with swollen joints | affected by SLE | arthritis at baseline |
| Hypothetical | Hypothetical | Composite | Hypothetical | | Composite | | | 9. | Composite | | | | Composite | | | Hypothetical | o v | | | Composite | Î | | |
| Prednisone (or equivalent) dose, change from | paseline | | TJC, change from | | | | | | >50% Reduction in | TJC | | | | | | SJC, change from | baseline | | | | | | |
| | | | TJC | | | | | | | | | | | | | SJC | | | | | | | |

LY3361237

| Exploratory | Exploratory | Exploratory | Exploratory | Exploratory | Exploratory | Exploratory | Exploratory |
|---|---|---|---|---|---|---|---|
| Logistic Regression with NRI Fisher's Exact Test with NRI Logistic Regression with NRI NRI | NRI<br>linear regression | linear regression with BOCF | linear regression | linear regression | Linear regression with<br>BOCF | Fisher's Exact Test | linear regression |
| LY3471851 vs Placebo at postbaseline visits in the treatment period LY3471851 vs Placebo at postbaseline visits in the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period |
| mITT – Patients with swollen joints affected by SLE arthritis at baseline mITT – Patients with ≥8 SJC at baseline | mITT | mITT | mITT – Patients<br>with elevated anti-<br>dsDNA level (>120<br>IU/mL) | mITT – Patients<br>with low C3 level at<br>baseline | mITT – Patients<br>with low C3 level at<br>baseline | mITT – Patients<br>with low C3 at<br>baseline | mITT – Patients<br>with low C4 level at<br>baseline |
| Composite<br>Composite | Hypothetical | Composite | Hypothetical | Hypothetical | Composite | Composite | Hypothetical |
| ≥50% Reduction in SJC | Anti-dsDNA,<br>change from<br>baseline | | | C3 level, change<br>from baseline | | Normal/high C3<br>level | C4 level, change<br>from baseline |
| | Serologic<br>Markers of<br>SLE | | | | | | |

LY3361237

| | | Composite | mITT – Patients<br>with low C4 level at<br>baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | linear regression with BOCF | Exploratory |
|---|---|---|---|---|---|---|
| | Normal/high C4<br>level | Composite | mITT – Patients<br>with low C4 at<br>baseline | LY3471851 vs Placebo<br>at postbaseline visits in<br>the treatment period | Fisher's Exact Test | Exploratory |
| | Time to first flare | Hypothetical | mITT | LY3471851 vs Placebo<br>during the treatment | Cox regression | Exploratory |
| | | (censored at | | period | Kaplan-Meier plot | |
| | | the time of | | | | |
| | | of concomitant | | | | |
| | | medication | | | | |
| | | rules if flare | | | | |
| | | not occurred | | | | |
| | | beforehand) | | | | |
| Severe<br>Flare | Time to first severe | Hypothetical | mITT | LY3471851 vs Placebo | Cox regression | Exploratory |
| | | (censored at | | period | Kaplan-Meier plot | |
| | | the time of | | | | |
| | | first violation | | | | |
| | | of concomitant | | | | |
| | | medication | | | | |
| | | rules if flare | | | | |
| | | not occurred | | | | |
| | | beforehand) | | | | |
| SLICC | SLICC Damage | Composite | mITT | LY3471851 vs Placebo | linear regression | Exploratory |
| Damage | Index, change from | | | at postbaseline visits in | | |
| Index | baseline | | | the treatment period | | |

intent-to-treat; NRI = non-responder imputation; PCS = Physical Component Summary; PGA = Physician's Global Assessment; SF = Short Form; SJC = Erythematosus Disease Area and Severity Index; LLDAS = Lupus Low Disease Activity State; MCS = Mental Component Summary; mITT = modified Swollen Joint Count; SLE = systemic lupus erythematosus; SLEDAI-2K = Systemic Lupus Erythematosus Disease Activity Index 2000; SLEDAI-4 = a >4-point reduction in SLEDAI-2K score from baseline; SLICC = Systemic Lupus Erythematosus International Collaborating Clinics; SRI-4 = Systemic Abbreviations: Anti-dsDNA = anti-double stranded deoxyribonucleic acid; BICLA = British Isles Lupus Assessment Group-based Composite Lupus Assessment; BILAG = British Isles Lupus Assessment Group - 2004; BOCF = baseline observation carried forward; CLASI = Cutaneous Lupus Lupus Erythematosus Responder Index-4; TJC = Tender Joint Count.

# 6.3. Appendix 3: SLEDAI-2K

The total SLEDAI score is a weighted sum of those questions that have been answered as "present" on the CRF. The weights are listed below. For example, if a patient's CRF was marked present on psychosis, arthritis and rash then their score would be 8+4+2=14.

For the SLEDAI questionnaire, if any, but not all, of the 24 item scores is missing then impute a score of 0 for the missing item(s) when calculating the total score. In addition, any item with missing data will be imputed as 'not present' for any other analyses if at least one of the 24 items is nonmissing. If all 24 item scores are missing, then the total score will be missing, as well as any other analysis by organ system or individual descriptor.

| Weight | SLEDAI<br>SCORE | Descriptor | Definition |
|---|---|---|---|
| 8 | 8 | _ Seizure | Recent onset, exclude metabolic, infectious or drug causes. |
| 8 | | _ Psychosis | Altered ability to function in normal activity due to severe disturbance in the perception of reality. Include hallucinations, incoherence, marked loose associations, impoverished thought content, marked illogical thinking, bizarre, disorganized, or catatonic behavior. Exclude uremia and drug causes. |
| 8 | - | Organic brain syndrome | Altered mental function with impaired orientation, memory, or other intellectual function, with rapid onset and fluctuating clinical features, inability to sustain attention to environment, plus at least 2 of the following: perceptual disturbance, incoherent speech, insomnia or daytime drowsiness, or increased or decreased psychomotor |
| 8 | 6 | Visual disturbance | activity. Exclude metabolic, infectious, or drug causes. Retinal changes of SLE. Include cytoid bodies, retinal hemorrhages, scrous exudate or hemorrhages in the choroid, or optic neuritis. Exclude hypertension, infection, or drug causes. |
| 8 | | Cranial nerve disorder | New onset of sensory or motor neuropathy involving cranial nerves. |
| 8 | N <del>a</del> | _ Lupus headachc | Severe, persistent headache; may be migrainous, but must be nonresponsive to narcotic analgesia. |
| 8 | | _ CVA | New onset of cerebrovascular accident(s). Exclude arteriosclerosis. |
| 8 | /38 | _ Vasculitis | Ulceration, gangrene, tender finger nodules, periungual infarction, splinter hemorrhages, or biopsy or angiogram proof of vasculitis. |
| 4 | · | _ Arthritis | ≥ 2 joints with pain and signs of inflammation (i.e., tendemess, swelling or effusion). |
| 4 | | _ Myositis | Proximal muscle aching/weakness, associated with elevated creatine phosphokinase/aldolase or electromyogram changes or a biopsy showing myositis. |
| 4 | | _ Urinary casts | Heme-granular or red blood cell casts. |
| 4 | 10. 000.000.00 | Hematuria | >5 red blood cells/high power field. Exclude stone, infection or other cause. |
| 4 | | _ Proteinuria | >0.5 gram/24 hours |
| 4 | | | >5 white blood cells/high power field. Exclude infection. |
| | (6)<br>Y <u>C ROWSON</u> | | Inflammatory type rash. |
| 2 | 0 | Alopecia | Abnormal, patchy or diffuse loss of hair. |
| 2<br>2<br>2 | | Mucosal ulcers | Oral or nasal ulcerations. |
| 2 | | _ Pleurisy | Pleuritic chest pain with pleural rub or effusion, or pleural thickening. |
| 2 | | Pericarditis | Pericardial pain with at least 1 of the following: rub, effusion, or electrocardiogram or echocardiogram confirmation. |
| 2 | | Low complement | Decrease in CH50, C3, or C4 below the lower limit of normal for testing laboratory |
| 2 | 108 | Increased DNA binding | Increased DNA binding by Farr assay above normal range for testing laboratory. |
| 1 | 0.5 | Fever | >38°C. Exclude infectious cause. |
| î | ( <del>)</del> | _ Thrombocytopenia | <100,000 platelets / x109/L, exclude drug causes. |
| Ī | 3.1 | Leukopenia | < 3,000 white blood cells / x109/L, exclude drug causes. |

TOTAL SLEDAI SCORE For the purposes of analyses by organ system, the following list shows what descriptors are part of each organ system:

- Central Nervous System: Seizure, Psychosis, Organic Brain Syndrome, Visual Disturbance, Cranial Nerve Disorder, Lupus Headache, CVA
- 2. Vascular: Vasculitis
- 3. Musculoskeletal: Arthritis, Myositis
- 4. Renal: Urinary Casts, Hematuria, Proteinuria, Pyuria
- 5. Mucocutaneous: Rash, Alopecia, Mucosal Ulcers
- 6. Cardiovascular and Respiratory: Pleurisy, Pericarditis
- 7. Immunologic: Low complement, Increased DNA Binding
- 8. Constitutional: Fever
- 9. Hematologic: Thrombocytopenia, Leukopenia

## 6.4. Appendix 4: BILAG 2004

The BILAG 2004 index is a validated global disease activity index designed on the basis of the physician's intent-to-treat, focusing on changes in disease manifestations (not present, improving, same, worse, or new) occurring in the last 4 weeks compared with the previous 4 weeks. The instrument assesses 97 clinical signs, symptoms, and laboratory parameters across 9 organ system domains: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal, and hematology.

For BILAG, any item that appears 'Not done' will be assumed to be 'Not present'. Any missing data will be assumed to also be 'Not present' if at least there is a nonmissing item in the whole questionnaire.

- The BILAG A disease activity score is severe disease activity requiring high-dosage oral or intravenous corticosteroids, immunomodulators, or high-dosage anticoagulation along with high-dosage corticosteroids or immunomodulators.
- The BILAG B disease activity score is moderate disease activity requiring low-dosage oral corticosteroids, intramuscular or intra-articular corticosteroid injections, topical corticosteroids or immunomodulators, antimalarials, or symptomatic therapy.
- The BILAG C corresponds to stable, mild disease.
- The BILAG D is inactive disease that was active previously.
- The BILAG E indicates the system was never involved.

#### Calculation of the BILAG A and B Disease Activity Scores for Each Domain

#### Constitutional

#### Category A:

Pyrexia recorded as 2 (same), 3 (worse), or 4 (new), and

Any 2 or more of the following recorded as 2 (same), 3 (worse), or 4 (new):

Weight loss

Lymphadenopathy/splenomegaly

Anorexia

#### Category B:

Pyrexia recorded as 2 (same), 3 (worse), or 4 (new), or

Any 2 or more of the following recorded as 2 (same), 3 (worse), or 4 (new):

Weight loss

Lymphadenopathy/splenomegaly

Anorexia

but do not fulfill criteria for Category A

#### Category C

Pyrexia recorded as 1 (improving) or

One or more of the following recorded as >0:

Weight loss

Lymphadenopathy/Splenomegaly

Anorexia

but does not fulfill criteria for category A or B

#### Category D

Previous involvement

#### Category E

No previous involvement

#### **MUCOCUTANEOUS**

#### Category A

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Skin eruption - severe

Angio-oedema - severe

Mucosal ulceration - severe

Panniculitis/Bullous lupus - severe

Major cutaneous vasculitis/thrombosis

#### Category B

Any Category A features recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Skin eruption - mild

Panniculitis/Bullous lupus - mild

Digital infarcts or nodular vasculitis

Alopecia - severe

#### Category C

Any Category B features recorded as 1 (improving) or

Any of the following recorded as >0:

Angio-oedema - mild

Mucosal ulceration - mild

Alopecia - mild

Periungual erythema/chilblains

Splinter haemorrhages

#### Category D

Previous involvement

#### Category E

No previous involvement

#### **NEUROPSYCHIATRIC**

#### Category A

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Aseptic meningitis

Cerebral vasculitis

Demyelinating syndrome

Myelopathy

Acute confusional state

Psychosis

Acute inflammatory demyelinating polyradiculoneuropathy

Mononeuropathy (single/multiplex)

Cranial neuropathy

Plexopathy

Polyneuropathy

Status epilepticus

Cerebellar ataxia

### Category B

Any Category A features recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Seizure disorder

Cerebrovascular disease (not due to vasculitis)

Cognitive dysfunction

Movement disorder

Autonomic disorder

Lupus headache - severe unremitting

Headache due to raised intracranial hypertension

#### Category C

Any Category B features recorded as 1 (improving)

#### Category D

Previous involvement

#### Category E

No previous involvement

#### **MUSCULOSKELETAL**

#### Category A

Any of the following recorded as 2 (same), 3 (worse) or 4 (new):

Severe Myositis

Severe Arthritis

#### Category B

Any Category A features recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Mild Myositis

Moderate Arthritis/Tendonitis/Tenosynovitis

#### Category C

Any Category B features recorded as 1 (improving) or

Any of the following recorded as >0:

Mild Arthritis/Arthralgia/Myalgia

#### Category D

Previous involvement

#### Category E

No previous involvement

#### CARDIORESPIRATORY

#### Category A

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Myocarditis/Endocarditis + Cardiac failure

Arrhythmia

New valvular dysfunction

Cardiac tamponade

Pleural effusion with dyspnoea

Pulmonary haemorrhage/vasculitis

Interstitial alveolitis/pneumonitis

Shrinking lung syndrome

**Aortitis** 

Coronary vasculitis

# Category B

Any Category A features recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Pleurisy/Pericarditis

Myocarditis - mild

#### Category C

Any Category B features recorded as 1 (improving)

#### Category D

Previous involvement

#### Category E

No previous involvement

# **GASTROINTESTINAL**

#### Category A

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Peritonitis

Lupus enteritis/colitis

Intestinal pseudo-obstruction

Acute lupus cholecystitis

Acute lupus pancreatitis

#### Category B

Any Category A feature recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Abdominal serositis and/or ascites

Malabsorption

Protein losing enteropathy

Lupus hepatitis

#### Category C

Any Category B features recorded as 1 (improving)

#### Category D

Previous involvement

#### Category E

No previous involvement

#### **OPHTHALMIC**

#### Category A

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Orbital inflammation/myositis/proptosis

Keratitis - severe

Posterior uveitis/retinal vasculitis - severe

Scleritis - severe

Retinal/choroidal vaso-occlusive disease

Optic neuritis

Anterior ischaemic optic neuropathy

#### Category B

Any Category A features recorded as 1 (improving) or

Any of the following recorded as 2 (same), 3 (worse), or 4 (new):

Keratitis - mild

Anterior uveitis

Posterior uveitis/retinal vasculitis - mild

Scleritis - mild

#### Category C

Any Category B features recorded as 1 (improving) or

Any of the following recorded as >0:

**Episcleritis** 

Isolated cotton-wool spots (cytoid bodies)

#### Category D

Previous involvement

#### Category E

No previous involvement

#### RENAL

#### Category A

Two or more of the following providing 1, 4, or 5 is included:

1. Deteriorating proteinuria (severe) defined as

- a. urine dipstick increased by ≥2 levels (used only if other methods of urine protein estimation not available); or
- b. 24-hour urine protein >1 g that has not decreased (improved) by 25%; or
- c. urine protein-creatinine ratio >100 mg/mmol that has not decreased (improved) by 25%; or
- d. urine albumin-creatinine ratio >100 mg/mmol that has not decreased (improved) by 25%.
- 2. Accelerated hypertension.
- 3. Deteriorating renal function (severe) defined as
  - a. plasma creatinine >130 mol/L and having risen to >130% of previous value; or
  - b. GFR <80 mL/min per 1.73 m<sup>2</sup> and having fallen to <67% of previous value; or
  - c. GFR <50 mL/min per 1.73 m<sup>2</sup> and last time was > 50 ml/min per 1.73 m<sup>2</sup> or was not measured.
- 4. Active urinary sediment
- 5. Histological evidence of active nephritis within last 3 months
- 6. Nephrotic syndrome

#### Category B

One of the following:

- 1. One of the Category A features
- 2. Proteinuria (that has not fulfilled Category A criteria)
  - a. urine dipstick which has risen by 1 level to at least 2+ (used only if other methods of urine protein estimation not available); or
  - b. 24-hour urine protein ≥0.5 g that has not decreased (improved) by 25%; or
  - c. urine protein-creatinine ratio ≥50 mg/mmol that has not decreased (improved) by 25%; or
  - d. urine albumin-creatinine ratio ≥50 mg/mmol that has not decreased (improved) by 25%
- 3. Plasma creatinine > 130 mol/L and having risen to ≥115% but ≤130% of previous value.

#### Category C

One of the following:

1. Mild/Stable proteinuria defined as

- a. urine dipstick ≥1+ but has not fulfilled criteria for Category A and B (used only if other methods of urine protein estimation not available); or
- b. 24-hour urine protein >0.25 g but has not fulfilled criteria for Category A and B; or
- c. urine protein-creatinine ratio >25 mg/mmol but has not fulfilled criteria for Category A and B; or
- d. urine albumin-creatinine ratio >25 mg/mmol but has not fulfilled criteria for Category A and B
- 2. Rising blood pressure (providing the recorded values are >140/90 mm Hg) which has not fulfilled criteria for Category A and B, defined as
  - a. systolic rise of ≥30 mm Hg; and
  - b. diastolic rise of ≥15mm Hg

#### Category D

Previous involvement

#### Category E

No previous involvement

Note: although albumin-creatinine ratio and protein-creatinine ratio are different, we use the same cut- off values for this index.

#### HEMATOLOGICAL

#### Category A

TTP recorded as 2 (same), 3 (worse), or 4 (new) or

#### Any of the following:

Haemoglobin <8 g/dLWhite cell count  $<1.0 \times 10^9/\text{L}$ Neutrophil count  $<0.5 \times 10^9/\text{L}$ Platelet count  $<2.5 \times 10^9/\text{L}$ 

#### Category B

#### TTP recorded as 1 (improving) or

#### Any of the following:

Haemoglobin 8 - 8.9 g/dLWhite cell count  $1 - 1.9 \times 10^9/\text{L}$ Neutrophil count  $0.5 - 0.9 \times 10^9/\text{L}$ Platelet count  $25 - 49 \times 10^9/\text{L}$ Evidence of active haemolysis

#### Category C

Any of the following:

Haemoglobin 9 - 10.9 g/dLWhite cell count  $2 - 3.9 \times 10^9 \text{/L}$ Neutrophil count  $1 - 1.9 \times 10^9 \text{/L}$ Lymphocyte count  $<1.0 \times 10^9 \text{/L}$ Platelet count  $50 - 149 \times 10^9 \text{/L}$ Isolated Coombs' test positive

#### Category D

Previous involvement

#### Category E

No previous involvement

#### **Numerical Categorization for BILAG A-E**

For each organ system domain, BILAG 2004 numeric score of A to E will be assigned according to the following rule (Yee et al. 2010)

- BILAG A disease activity score = 12 points
- BILAG B disease activity score = 8 points
- BILAG C disease activity score = 1 point
- BILAG D disease activity score = 0 points
- BILAG E disease activity score = 0 points

For each complete BILAG assessment, the points score from each of the nine BILAG organ system domains will be summed to obtain a BILAG 2004 numeric score. The numeric score will only be calculated if each of the 9 disease activity scores are nonmissing.

# 6.5. Appendix 5: Joint Assessment

The 28 joints will be evaluated for tenderness and 28 joints will be evaluated for swelling (hips are excluded for swelling) at the specified visits as shown in the schedule of events of the protocol. The 28 joint count will be performed at Week 0 (V2/baseline), Week 2 (V4) to Week 24 (V14), end of treatment, and at follow-up visit.

The following joint count imputation rules will be applied.

- 1. Joints that had any of the following procedures or disease conditions that occur at the screening (Visit 1), up to and including baseline (Visit 2), will be imputed as follows:
  - a. Arthroplasty, fusion, synovectomy, ankylosis, amputation, injury, fracture, infection and other condition: these will be considered "nonevaluable" from baseline up to end of the study. Joints that include "nonevaluable" joints will be prorated from baseline up to end of the study. For example, the swollen joint count score for 6 swollen plus 2 "nonevaluable" joints is calculated as [6/(28-2)]\*28 = 6.46.
  - b. Injection and other procedure: joints that have received intra-articular and bursal injections will be collected in the data but set to painful/tender or swollen after the injection for 6 months (up to Week 24 (V15) [Visit 9]).
- Joints that had any of the following procedures or disease conditions that occur postbaseline (any time during treatment with the study drugs) will be imputed as follows:
  - a. Amputation: amputation that occurs postbaseline will be considered "nonevaluable" from the visit after amputation up to end of the study. Joints that include "nonevaluable" joints will be pro-rated from the visit after amputation up to end of the study. For example, the swollen joint count score for 6 swollen plus 2 "nonevaluable" joints is calculated as [6/(28-2)]\*28 = 6.46.
  - b. Arthroplasty, fusion, synovectomy, and ankylosis: if any of these procedures occur postbaseline, joints will be set to tender and swollen from the visit after the procedure up to the end of the study.
  - c. Infection, injury, and fracture or other condition: if any of these conditions occur postbaseline, joints will be set to tender and swollen from the visit after the condition until the condition is resolved.
  - d. Injection and other procedure: joints that have received intra-articular and bursal injections postbaseline will be collected in the data but set to tender and swollen after the injection for 6 months or the end of the study (whichever comes first).

The number of tender and swollen joints will be calculated by summing all joints respectively. For patients who have an incomplete set of joints evaluated, the joint count will be adjusted to a 28-joint count for tenderness and a 28-joint count for swelling by dividing the number of affected joints by the number of evaluated joints and multiplying by 28 for tenderness and 28 for swelling.

# 6.6. Appendix 6: SLICC/ARC Damage Index

The total score is a simple sum of all 39 items on the CRF. Note that while most items are scored either 0 (not present) or 1 (present), there are some items that are weighted heavier. Note for example that the following items can have a response of either 0, 1 or 2 on the CRF. If "2" is selected that is what should be included in the sum

- Cerebrovascular accident.
- myocardial infarction,
- significant tissue loss
- infarction or resection of bowel
- avascular necrosis
- malignancy

Also note for end stage renal failure, it is either 0 (not present) or 3 (present). If it is present, then the score of 3 is added to the total.

# 6.7. Appendix 7: Corticosteroid Conversion

All corticosteroid doses need to be converted to prednisone equivalent doses (as detailed in Section 6.8). If additional conversion factors are required, these will be added to the table below in a statistical analysis plan amendment prior to database lock.

The following table should be used for converting nonprednisone medications to prednisone equivalent:

Multiply the dose of the corticosteroid taken by the patient (in milligrams) in Column 1 by the conversion factor in Column 2 to get the equivalent dose of prednisone (in milligrams). Example: Patient is taking 16 mg of methylprednisolone po daily. To convert to prednisone: 16 mg methylprednisolone  $\times 1.25 = 20 \text{ mg}$  prednisone. 16 mg of methylprednisolone po daily is equivalent to 20 mg of prednisone po daily.

Table APP.7.1. Corticosteroid Conversion

| Column 1 | Column 2 |
|---|---|
| Corticosteroid Preferred Term | Conversion factor for converting to an equivalent prednisone dose |
| Prednisone | 1 |
| Prednisone acetate | 1 |
| Prednisolone | 1 |
| Prednisolone acetate | 1 |
| Prednisolone sodium phosphate | 1 |
| Methylprednisolone | 1.25 |
| Methylprednisolone acetate | 1.25 |
| Methylprednisolone sodium succinate | 1.25 |
| Triamcinolone | 1.25 |
| Triamcinolone acetonide | 1.25 |
| Triamcinolone hexacetonide | 1.25 |
| Cortisone | 0.2 |
| Cortisone acetate | 0.2 |
| Hydrocortisone | 0.25 |
| Hydrocortisone acetate | 0.25 |
| Hydrocortisone sodium succinate | 0.25 |
| Betamethasone | 6.25 |
| Betamethasone acetate | 6.25 |
| Betamethasone dipropionate | 6.25 |
| Betamethasone sodium phosphate | 6.25 |
| Dexamethasone | 6.25 |
| Dexamethasone acetate | 6.25 |
| Dexamethasone phosphate | 6.25 |
| Dexamethasone sodium phosphate | 6.25 |
| Paramethasone | 2.5 |
| Deflazacort | 0.83 |
| Celestona bifas | 6.25 |
| Depo-medrol med lidokain | 1.25 |
| Diprospan | 6.25 |
| Fluocortolone | 1 |
| Meprednisone | 1.25 |

#### 6.8. Appendix 8: Corticosteroid Management

Key elements of corticosteroid management in this study include the following:

- Enrolled participants are restricted to prednisone ≤20 mg per day (or equivalent) at randomization (Visit 2), having been on stable doses for at least 2 weeks prior to randomization.
- Following randomization, the dose of prednisone (or equivalent) should not be increased above the participant's background level (dose at baseline).
- Participants on ≥10 mg per day are required to taper their dose to taper their dose to
   10 mg per day by Week 12, and maintain a dose <10 mg to Week 24 to be considered responders.</li>
- Participants with intolerable or exacerbating disease are allowed access to standard of
  care therapy, including increasing the dose of prednisone (or equivalent). Such
  participants are allowed to remain in the study but will be permanently discontinued
  from study intervention (see the Master Protocol IMMA [Section 7.1]).

# 6.9. Appendix 9: List of MedDRA Preferred Terms for Potential Opportunistic Infections

Table APP.9.1. MedDRA Preferred Terms for POI

| Category | Potential Opportunistic<br>Infection | Preferred Term<br>(MedDRA Version<br>22.1) | Preferred Term<br>Code | Lilly Defined<br>Classification |
|---|---|---|---|---|
| Mycobacterial/ | Nocardiosis (II) | Nocardia sepsis | 10064952 | Narrow |
| Actino | 1.50 | Nocardiosis | 10029444 | |
| | | Nocardia test positive | 10070131 | Broad |
| Mycobacterial/<br>Actino | Nontuberculous<br>mycobacterium disease | Atypical mycobacterial infection | 10061663 | Narrow |
| | (II) | Atypical mycobacterial lower respiratory tract infection | 10075026 | |
| | | Atypical mycobacterial lymphadenitis | 10003755 | |
| | | Atypical mycobacterium pericarditis | 10055036 | |
| | | Atypical mycobacterial pneumonia | 10071075 | |
| | | Borderline leprosy | 10006029 | |
| | | Bovine tuberculosis | 10006049 | 1 |
| | | Indeterminate leprosy | 10021700 | |
| | | Leprosy | 10024229 | 1 |
| | | Lepromatous leprosy | 10024227 | |
| | | Mycobacterial infection | 10062207 | 1 |
| | | Mycobacterial peritonitis | 10073514 | |
| | | Mycobacterium<br>abscessus infection | 10064789 | |
| | | Mycobacterium avium complex immune restoration disease | 10058449 | |
| | | Mycobacterium avium complex infection | 10058806 | |
| | | Mycobacterium chelonae infection | 10071401 | |
| | | Mycobacterium<br>fortuitum infection | 10049659 | |
| | | Mycobacterium kansasii infection | 10028447 | |
| | | Mycobacterium<br>marinum infection | 10028452 | |
| | | Mycobacterium ulcerans infection | 10066289 | |

| | ř | | 10055001 | |
|---|---|---|---|---|
| | | Superinfection | 10075381 | |
| | | mycobacterial | 10044550 | - |
| | | Tuberculoid leprosy | 10044729 | 4 |
| | | Type 1 lepra reaction | 10070516 | 4 |
| | | Type 2 lepra reaction | 10070517 | |
| | | Atypical mycobacterium | 10070326 | Broad |
| | | test positive | | |
| | | Mycobacterial disease | 10075025 | |
| | | carrier | | |
| | | Mycobacterium leprae | 10070324 | |
| | | test positive | | |
| | | Mycobacterium test | 10070407 | |
| | | Mycobacterium test | 10070323 | |
| | | positive | Emergentation resists | |
| | | Ureaplasmal | 10081280 | 1 |
| | | ulvovaginitis | | |
| Mycobacterial/ | Tuberculosis (I) | Adrenal gland | 10001358 | Narrow |
| Actino | | tuberculosis | 200 TABLE TO THE TOTAL TO THE SECOND | |
| | | Bone tuberculosis | 10056377 | 1 |
| | | Choroid tubercles | 10008779 | - |
| | | | and or the second second second | - |
| | | Congenital tuberculosis | 10010657 | _ |
| | | Conjunctivitis | 10010754 | |
| | | tuberculous | | _ |
| | | Cutaneous tuberculosis | 10011684 | _ |
| | | Disseminated Bacillus | 10076666 | |
| | | Calmette-Guerin | | |
| | | infection | | _ |
| | | Disseminated | 10013453 | |
| | | tuberculosis | | |
| | | Ear tuberculosis | 10014027 | |
| | | Epididymitis | 10015004 | |
| | | tuberculous | | |
| | | Extrapulmonary | 10064445 | |
| | | tuberculosis | | 1 |
| | | Female genital tract | 10061150 | |
| | | tuberculosis | | 1 |
| | | Immune reconstitution | 10072797 | |
| | | inflammatory syndrome | | |
| | | associated tuberculosis | | _ |
| | | Intestinal tuberculosis | 10075268 | |
| | | Joint tuberculosis | 10056367 | |
| | | Lupus vulgaris | 10025143 | 1 |
| | | Lymph node | 10025183 | 1 |
| | | tuberculosis | | |
| | | Male genital tract | 10061234 | 1 |
| | | tuberculosis | | |
| | | Meningitis tuberculous | 10027259 | 1 |
| | l . | The state of the s | 1002/202 | L |

| | 0 1 1 | 10000000 | 9 |
|--|---|---|---|
| | Oesophageal | 10030200 | |
| | tuberculosis | 10076970 | |
| | Oral tuberculosis | 10076879 | |
| | Pericarditis tuberculous | 10055069 | |
| | Peritoneal tuberculosis | 10053583 | |
| | Prostatitis tuberculous | 10064743 | |
| | Pulmonary tuberculoma | 10066927 | |
| | Pulmonary tuberculosis | 10037440 | |
| | Renal tuberculosis | 10038534 | |
| | Salpingitis tuberculous | 10039463 | |
| | Silicotuberculosis | 10068876 | |
| | Spleen tuberculosis | 10041640 | |
| | Thyroid tuberculosis | 10043774 | |
| | Tuberculoma of central | 10052883 | |
| | nervous system | | |
| | Tuberculosis | 10044755 | |
| | Tuberculosis bladder | 10044758 | |
| | Tuberculosis | 10061390 | |
| | gastrointestinal | | |
| | Tuberculosis liver | 10058120 | |
| | Tuberculosis of central | 10061391 | |
| | nervous system | W | |
| | Tuberculosis of eye | 10044819 | |
| | Tuberculosis of | 10044828 | |
| | genitourinary system | N. Strongella, Box V. C. C. C. | |
| | Tuberculosis of | 10044846 | |
| | intrathoracic lymph | | |
| | nodes | **** | |
| | Tuberculosis of | 10044965 | |
| | peripheral lymph nodes | 10045026 | |
| | Tuberculosis ureter | 10045026 | |
| | Tuberculous abscess | 10052884 | |
| | central nervous system Tuberculous | 10071550 | |
| | endometritis | 10071559 | |
| | Tuberculous laryngitis | 10045072 | |
| | Tuberculous pleurisy | 10045104 | |
| | Tuberculous Tuberculous | 10043104 | |
| | tenosynovitis | 10039101 | |
| | Interferon gamma | 10073542 | Broad |
| | release assay | 100/3342 | Diouci |
| | Interferon gamma | 10072866 | |
| | release assay positive | 100/2000 | |
| | Mycobacterium | 10070472 | |
| | tuberculosis complex | 20010112 | |
| | test | | |
| | Mycobacterium<br>tuberculosis complex<br>test positive | 10070325 | |
|---|---|---|---|
| | Tuberculid | 10044725 | 1 |
| | Tuberculin test | | 1 |
| | Tuberculin test false negative | 10074840 | |
| | | 10044728 | |
| Bartonellosis | | 10003971 | Narrow |
| (disseminated disease | Trench fever | 10044582 | |
| only) (V) | Bartonella test | 10075209 | Broad |
| 25.Col355 B | Bartonella test positive | | |
| | Bartonellosis | | |
| | | The state of the s | |
| Campylobacteriosis | | 10070681 | Narrow |
| 9112.00 | The state of the s | 10076769 | Broad |
| (V) | Campylobacter<br>gastroenteritis | 10007048 | |
| | Campylobacter infection | 10051226 | 1 |
| | Campylobacter test positive | 10070025 | |
| Legionellosis (II) | Legionella infection | 10061266 | Narrow |
| | Pneumonia legionella | 10035718 | |
| | Pontiac fever | 10054161 | |
| | Legionella test | 10070410 | Broad |
| | Legionella test positive | 10070092 | |
| Listeria monocytogenes | Listeria encephalitis | 10054116 | Narrow |
| (invasive disease only) | Listeria sepsis | 10063085 | |
| (II) | Meningitis listeria | 10027248 | |
| | Listeria test | 10075707 | Broad |
| | Listeria test positive | 10070094 | |
| | Listeriosis | 10024641 | |
| Salmonellosis (invasive | Aortitis salmonella | 10074937 | Narrow |
| disease only) (II) | Arthritis salmonella | 10003271 | |
| | Meningitis salmonella | 10027254 | |
| | Osteomyelitis<br>salmonella | 10031262 | |
| | Paratyphoid fever | 10033971 | |
| | | 10033971<br>10035733 | - |
| | Paratyphoid fever | | |
| | Paratyphoid fever<br>Pneumonia salmonella | 10035733 | |
| | Paratyphoid fever<br>Pneumonia salmonella<br>Salmonella bacteraemia<br>Salmonella sepsis | 10035733<br>10058924 | |
| | Paratyphoid fever Pneumonia salmonella Salmonella bacteraemia Salmonella sepsis Typhoid fever | 10035733<br>10058924<br>10058878 | Broad |
| | Paratyphoid fever<br>Pneumonia salmonella<br>Salmonella bacteraemia<br>Salmonella sepsis | 10035733<br>10058924<br>10058878<br>10045275 | Broad |
| | Paratyphoid fever Pneumonia salmonella Salmonella bacteraemia Salmonella sepsis Typhoid fever Salmonella test positive | 10035733<br>10058924<br>10058878<br>10045275<br>10070127 | Broad |
| | (disseminated disease only) (V) Campylobacteriosis (invasive disease only) (V) Legionellosis (II) Listeria monocytogenes (invasive disease only) (II) | tuberculosis complex test positive Tuberculid Tuberculin test Tuberculin test false negative Tuberculin test positive Bartonellosis (disseminated disease only) (V) Bartonella test Bartonella test Bartonella test Bartonella test positive Cat scratch disease Peliosis hepatis Splenic peliosis Campylobacter sepsis (invasive disease only) (V) Campylobacter colitis Campylobacter gastroenteritis Campylobacter infection Campylobacter infection Campylobacter test positive Legionella infection Pneumonia legionella Pontiac fever Legionella test positive Listeria encephalitis Listeria encephalitis Listeria test positive Listeria test Listeria test Listeria test positive Listeriosis Salmonellosis (invasive disease only) (II) Arthritis salmonella Meningitis salmonella | tuberculosis complex test positive Tuberculid |

| | Shigellosis (invasive | Shigella infection | 10054178 | Broad |
|---|---|---|---|---|
| | disease only) (V) | Shigella test positive | 10070129 | 101111111111111111111111111111111111111 |
| | Vibriosis (invasive | Gastroenteritis vibrio | 10017917 | Broad |
| | disease due to $V$ . | Vibrio test positive | 10070161 | 0 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| | vulnificus) (V) | None | | Narrow |
| | Infective Pneumonia | Pneumonia | 10079866 | Narrow |
| | SMQ | acinetobacter | | |
| | | Pneumonia proteus | 10079867 | |
| | | Pneumonia serratia | 10079868 | |
| Fungal | Aspergillosis (invasive | Aspergillosis oral | 10003489 | |
| | disease only) (II) | Cerebral aspergillosis | 10051597 | |
| | , | Meningitis aspergillus | 10073245 | |
| | | Oro-pharyngeal<br>aspergillosis | 10053029 | |
| | | Aspergillus infection | 10074171 | |
| | | Aspergillus test | 10070450 | |
| | | Aspergillus test positive | 10070448 | |
| | | Bronchopulmonary | 10006473 | |
| | | aspergillosis | 10000175 | |
| | | Sinusitis aspergillus | 10051016 | |
| | Blastomycosis (IV) | Blastomycosis | 10005098 | Narrow |
| | Diagram (11) | Epididymitis | 10015001 | |
| | | blastomyces | | |
| | | Osteomyelitis | 10031255 | |
| | | blastomyces | | |
| | | Pneumonia blastomyces | 10035671 | |
| | | None | 10000071 | Broad |
| | Candidiasis (invasive | Candida | 10059449 | Narrow |
| | disease, or oral not limited | endophthalmitis | | <u> </u> |
| | to the tongue) (II) | Candida osteomyelitis | 10064699 | |
| | 30 305 R.S. S. S. S. A. A. A. | Candida pneumonia | 10053158 | |
| | | Candida retinitis | 10068612 | |
| | | Candida sepsis | 10053166 | |
| | | Candida urethritis | 10081262 | |
| | | Candidiasis of trachea | 10064459 | |
| | | Cerebral candidiasis | 10078126 | |
| | | Endocarditis candida | 10014669 | |
| | | Gastrointestinal | 10017938 | |
| | | candidiasis | | |
| | | Hepatic candidiasis | 10049653 | |
| | | Hepatosplenic | 10051590 | |
| | | candidiasis | | |
| | | Meningitis candida | 10027205 | |
| | | Oesophageal candidiasis | 10030154 | |
| | | Oral candidiasis | 10030963 | |
| | | Oropharyngeal | 10050346 | |
| | | candidiasis | | |
| | | Peritoneal candidiasis | 10056562 | _ |

| | Splenic candidiasis | 10051725 | 3 |
|---|---|---|---|
| | Systemic candida | 10031723 | _ |
| | Bladder candidiasis | 10042938 | Broad |
| | Candida infection | 10038323 | Dioad |
| | | | - |
| | Candida test | 10070453 | - |
| | Candida test positive | 10070451 | _ |
| | Mucocutaneous | 10028080 | |
| | candidiasis <sup>1</sup> | | |
| | Respiratory moniliasis | 10038705 | |
| Coccidioidomycosis (II) | Coccidioides | 10054214 | Narrow |
| | encephalitis | | |
| | Coccidioidomycosis | 10009825 | |
| | Cutaneous | 10068747 | |
| | coccidioidomycosis | | |
| | Meningitis coccidioides | 10027207 | 03 |
| | None | | Broad |
| Cryptococcosis (II) | Cryptococcal cutaneous | 10054216 | Narrow |
| 987 VARIA | infection | | |
| | Cryptococcal fungaemia | 10067112 | |
| | Cryptococcosis | 10011490 | |
| | Disseminated | 10013439 | |
| | cryptococcosis | 4-48-6-3-4-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1-1 | |
| | Gastroenteritis | 10011485 | |
| | cryptococcal | | |
| | Meningitis cryptococcal | 10027209 | |
| | Neurocryptococcosis | 10068368 | |
| | Pneumonia cryptococcal | 10067565 | |
| | Cryptococcus test | 10070456 | Broad |
| | Cryptococcus test | 10070455 | Dioad |
| | positive | 10070433 | |
| Histoplasmosis (II) | Acute pulmonary | 10001027 | Narrow |
| Thstopiasmosis (II) | histoplasmosis | 10001027 | Nariow |
| | Chronic pulmonary | 10009115 | _ |
| | histoplasmosis | 10009113 | |
| | Endocarditis | 10014676 | - |
| | The state of the s | 10014676 | |
| | histoplasma | 10020141 | - |
| | Histoplasmosis | 10020141 | |
| | Histoplasmosis | 10049142 | |
| | cutaneous | | _ |
| | Histoplasmosis | 10020144 | |
| | disseminated | British - 200-200 | _ |
| | Meningitis histoplasma | 10027243 | |
| | Pericarditis histoplasma | 10034489 | |
| | Retinitis histoplasma | 10038912 | |
| | Presumed ocular | 10063664 | Broad |
| | histoplasmosis | | |
| | syndrome | | |
| | Microsporidia infection | | |

| | TORREST 10 1 78 829 1 8 | | | Broad |
|---|---|---|---|---|
| | Other invasive fungi: | Allescheriosis | 10001754 | Narrow |
| | Mucormycosis | Fusarium infection | 10051919 | |
| | (=zygomycosis) | Mucormycosis | 10028098 | |
| | [Rhizopus, Mucor, and | Scedosporium infection | 10059045 | |
| | Lichtheimia], | Pseudallescheria | 10061919 | |
| | Scedosporum/ | infection | | |
| | Pseudallescheria boydii, | Pseudallescheria sepsis | 10058973 | a |
| | Fusarium (II) | See "Non-specific<br>terms" below | | Broad |
| | Paracoccidioides | Paracoccidioides | 10061906 | Narrow |
| | infections (V) | infection | ************************************** | 5000000 M 50 M 5000 CO 11 |
| | The state of the s | None | | Broad |
| | Penicillium marneffei (V) | Penicillium infection | 10078580 | Narrow |
| | | None | | Broad |
| | Pneumocystis jirovecii (II) | Pneumocystis jirovecii infection | 10073756 | Narrow |
| | Pneumocystis jirovecii pneumonia | 10073755 | | |
| | | Blood beta-D-glucan | 10068725 | Broad |
| | | Blood beta-D-glucan | 10051795 | |
| | | abnormal | | |
| | | Blood beta-D-glucan | 10051793 | |
| | | increased | | |
| | | Gomori methenamine silver stain | 10075549 | |
| | 1 | Carbon monoxide | 10065906 | |
| | | diffusing capacity | | |
| | | decreased | | |
| | | Carbon monoxide | 10071738 | |
| | | diffusing capacity | 4 | |
| | | Pneumocystis test | 10070454 | |
| | | positive | | |
| | Sporothrix schenckii (V) | Cutaneous | 10011676 | Narrow |
| | | sporotrichosis | | |
| | | Sporotrichosis | 10041736 | - |
| cost la | 10 Annual Control of the Control of | None | | Taysons |
| Viral | TO COLOR OF THE CO | Cytomegalovirus | 10048843 | Narrow |
| | (V) | 3. 7 (4) 7 (4) | 1 | _ |
| | | Cytomegalovirus colitis | 10048983 | |
| | | Cytomegalovirus | 10049014 | |
| | | | 10040074 | - |
| | | | 100490/4 | |
| | | NAME OF TAXABLE PARTY. | 10040015 | $\dashv$ |
| | | enterocolitis | 10049013 | |
| | | Cytomegalovirus | 10049016 | - |
| | | gastritis | 10049010 | |
| Viral | Cytomegalovirus disease | Cutaneous sporotrichosis Sporotrichosis None Cytomegalovirus chorioretinitis Cytomegalovirus colitis Cytomegalovirus duodenitis Cytomegalovirus enteritis Cytomegalovirus | 10041736<br>10048843<br>10048983 | Broad |

| 8 | ľ | | 10051240 | 18 |
|---|---|---|---|---|
| | | Cytomegalovirus | 10051349 | |
| | | gastroenteritis | | _ |
| | | Cytomegalovirus | 10052817 | |
| | | gastrointestinal infection | | _ |
| | | Cytomegalovirus | 10075619 | |
| | | gastrointestinal ulcer | | |
| | | Cytomegalovirus | 10011830 | |
| | | hepatitis | | |
| | | Cytomegalovirus | 10011831 | |
| | | infection | | |
| | | Cytomegalovirus | 10011834 | |
| | | mononucleosis | | |
| | | Cytomegalovirus | 10065036 | |
| | | mucocutaneous ulcer | | |
| | | Cytomegalovirus | 10065621 | |
| | | myelomeningoradiculitis | The state of the s | |
| | | Cytomegalovirus | 10056261 | 1 |
| | | myocarditis | | |
| | | Cytomegalovirus | 10079095 | 1 |
| | | nephritis | | |
| | | Cytomegalovirus | 10049018 | 1 |
| | | oesophagitis | 10015010 | |
| | | Cytomegalovirus | 10049566 | - |
| | | pancreatitis | 10045500 | |
| | | Cytomegalovirus | 10056721 | 1 |
| | | pericarditis | 10030721 | |
| | | Cytomegalovirus | 10056262 | _ |
| | | syndrome | 10030202 | |
| | | Cytomegalovirus | 10051350 | - |
| | | urinary tract infection | 10031330 | |
| | | | 10058854 | - |
| | | Cytomegalovirus | 10038834 | |
| | | viraemia | 10040075 | - |
| | | Disseminated | 10049075 | |
| | | cytomegaloviral | | |
| | | infection | 10014505 | 4 |
| | | Encephalitis | 10014586 | |
| | | cytomegalovirus | 10005656 | 4 |
| | | Pneumonia | 10035676 | |
| | | cytomegaloviral | | |
| | | Cytomegalovirus test | 10061806 | Broad |
| | | Cytomegalovirus test | 10051620 | |
| | | positive | | |
| | HBV reactivation (IV) | None | | Narrow |
| | | Asymptomatic viral hepatitis | 10063838 | Broad |
| | | Chronic hepatitis B | 10008910 | 1 |
| | | HBV DNA polymerase | 10058937 | 1 |
| | | increased | 2000000 | |
| | I . | LIVI CUDE | I | 1 |

| | | Hepatitis B | 10019731 | |
|---|---|---|---|---|
| | | The second secon | 10019731 | - |
| | | Hepatitis B antigen | | 1 |
| | | Hepatitis B antigen | 10063411 | |
| | | positive | 10051160 | - |
| | | Hepatitis B core antigen | 10051160 | - |
| | | Hepatitis B core antigen | 10052328 | |
| | | positive | E-Service E-Service | - |
| | | Hepatitis B DNA assay | 10060027 | 4 |
| | | Hepatitis B DNA assay | 10060047 | |
| | | positive | | |
| | | Hepatitis B DNA | 10068379 | |
| | | increased | - | |
| | | Hepatitis B e antigen | 10050914 | |
| | | Hepatitis B e antigen | 10052329 | |
| | | positive | | ] |
| | | Hepatitis B reactivation | 10058827 | ] |
| | | Hepatitis B surface | 10050529 | |
| | | antigen | | |
| | | Hepatitis B surface | 10019742 | 1 |
| | | antigen positive | \$199-15000 (\$150 T) F) = 15000 T) | |
| | | Hepatitis B virus test | 10068415 | 1 |
| | | Hepatitis B virus test | 10070217 | 1 |
| | | positive | | |
| | | Hepatitis A | 10019780 | 1 |
| | | Hepatitis post | 10019791 | 1 |
| | | transfusion | 10015,51 | |
| | | Hepatitis viral | 10019799 | 1 |
| | | Withdrawal hepatitis | 10071220 | 1 |
| Viral | HCV progression (V) | None | 10071220 | Narrow |
| V II III | ine v progression (v) | Chronic hepatitis C | 10008912 | Broad |
| | | Hepatitis C | 10019744 | Dioad |
| | | Hepatitis C RNA | 10019744 | 1 |
| | | | | 1 |
| | | Hepatitis C RNA fluctuation | 10068727 | |
| | | ALCOHOLOGIC DESCRIPTION OF THE PROPERTY OF THE | 10069277 | 1 |
| | | Hepatitis C RNA | 10068377 | |
| | | increased | 10010750 | 1 |
| | | Hepatitis C RNA | 10019750 | |
| | | positive | 10060416 | 4 |
| | | Hepatitis C virus test | 10068416 | - |
| | | Hepatitis C virus test | 10070218 | |
| | | positive | | Transport |
| | Herpes simplex (IV) | Colitis herpes | 10051782 | Narrow |
| | | Eczema herpeticum | 10014197 | 4 |
| | | Gastritis herpes | 10051784 | 1 |
| | | Herpes oesophagitis | 10052330 | 1 |
| | | Herpes sepsis | 10058876 | ] |
| | | Herpes simplex colitis | 10074239 | |

| T | TT0222200.***** | 10010053 | 9 |
|---|---|---|---|
| | Herpes simplex | 10019953 | |
| | encephalitis | 10074240 | 1 |
| | Herpes simplex gastritis | 10074240 | 1 |
| | Herpes simplex hepatitis | 10067389 | - |
| | Herpes simplex | 10019956 | |
| | meningitis | | |
| | Herpes simplex | 10074247 | |
| | meningoencephalitis | 5-5-5-2-5-5-5 | |
| | Herpes simplex | 10074250 | |
| | meningomyelitis | | |
| | Herpes simplex | 10074252 | |
| | necrotising retinopathy | Bedrick and a participation | |
| | Herpes simplex oesophagitis | 10074242 | |
| | Herpes simplex | 10065046 | 1 |
| | pneumonia | 010000000000000000000000000000000000000 | |
| | Herpes simplex sepsis | 10074246 | 1 |
| | Herpes simplex visceral | 10019963 | 1 |
| | Meningitis herpes | 10027242 | 1 |
| | Meningoencephalitis | 10027242 | 1 |
| | herpetic | 1001/200 | |
| | Meningomyelitis herpes | 10074249 | |
| | Pneumonia herpes viral | 10074249 | 1 |
| | Genital herpes simplex | 10073931 | 1 |
| | Herpes dermatitis | 10062639 | 1 |
| | Herpes pharyngitis | 10066888 | |
| | Herpes simplex otitis | 10000888 | 1 |
| | externa | 10019939 | |
| | Herpes simplex | 10074244 | 1 |
| | pharyngitis | 100/4244 | |
| | | 10072020 | - |
| | Ophthalmic herpes<br>simplex | 10073938 | |
| | | 10026790 | 1 |
| | Proctitis herpes | 10036780 | 1 |
| | Kaposi's varicelliform | 10051891 | |
| | eruption Herpes simplex test | 10077060 | Broad |
| | | 10077969 | Broad |
| | positive | 10010049 | 1 |
| | Herpes simplex | 10019948 | 1 |
| | Herpes virus infection | 10019973 | 1 |
| | Nasal herpes | 10074936 | 1 |
| | Oral herpes | 10067152 | 1 |
| TT 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 2 | Genital herpes | 10018150 | 3.7 |
| Herpes zoster (any form) | Disseminated varicella | 10076667 | Narrow |
| (II) | zoster vaccine virus | | |
| | infection | 10014602 | - |
| | Encephalitis post | 10014603 | |
| | varicella | 10056510 | - |
| | Genital herpes zoster | 10072210 | ia . |

| 100 | | Herpes zoster | 10019974 | ia a |
|---|---|---|---|---|
| | | Herpes zoster cutaneous | 10074297 | 1 |
| | | disseminated | 100/425/ | |
| | | Herpes zoster | 10065038 | 1 |
| | | disseminated | 10003030 | |
| | | Herpes zoster infection | 10061208 | 1 |
| | | neurological | 10001200 | |
| | | Herpes zoster meningitis | 10074259 | 1 |
| | | Herpes zoster | 10074248 | 1 |
| | | meningoencephalitis | | |
| | | Herpes zoster | 10074251 | 1 |
| | | meningomyelitis | | |
| | | Herpes zoster | 10079327 | 1 |
| | | meningoradiculitis | of the third and the control of the | |
| | | Herpes zostemecrotising | 10074253 | 1 |
| | | retinopathy | | |
| | Ì | Herpes zoster oticus | 10063491 | ] |
| | | Herpes zoster | 10074245 | ] |
| | | pharyngitis | | |
| | | Necrotising herpetic | 10065119 | |
| | | retinopathy | | |
| | | Ophthalmic herpes | 10030865 | |
| | | zoster | | |
| | | Varicella | 10046980 | |
| | | Varicella keratitis | 10077496 | |
| | | Varicella post vaccine | 10063522 | |
| | | Varicella zoster gastritis | 10074241 | |
| | | Varicella zoster | 10074243 | |
| | | oesophagitis | | |
| | | Varicella zoster | 10074254 | |
| | | pneumonia | | |
| | | Varicella zoster virus | 10075611 | |
| | | infection | 1 | 1 |
| | | Herpes ophthalmic | 10062004 | |
| | | Varicella virus test | 10070444 | Broad |
| | | Varicella virus test | 10070214 | |
| | | positive | | |
| | Human Polyomavirus | BK virus infection | 10055181 | Narrow |
| | infection including BK | Human polyomavirus | 10057366 | |
| | virus disease and PVAN | infection | | 4 |
| | (V), and Progressive | JC virus granule cell | 10074361 | |
| | Multifocal | neuronopathy | 10000160 | 4 |
| | Leukoencephalopathy | JC virus infection | 10023163 | - |
| | (IV) | Polyomavirus-associated | 10065381 | |
| | | nephropathy | 1000000= | 4 |
| | | Progressive multifocal | 10036807 | |
| | | leukoencephalopathy | 1000050 | D 1 |
| | | JC virus test | 10068794 | Broad |

| | | Polyomavirus test | 10075038 | |
|---|---|---|---|---|
| | | Polyomavirus test<br>positive | 10070342 | |
| | Post-transplant<br>lymphoproliferative<br>disorder (EBV) (V) | Epstein-Barr virus<br>associated<br>lymphoproliferative<br>disorder | 10068349 | Narrow |
| | | Post-transplant<br>lymphoproliferative<br>disorder | 10051358 | |
| | | Epstein-Barr viraemia | 10065110 | Broad |
| | | Epstein-Barr virus<br>associated lymphoma | 10071441 | |
| | | Epstein-Barr virus infection | 10015108 | |
| | | Lymphoproliferative disorder | 10061232 | |
| | | Lymphoproliferative disorder in remission | 10061233 | |
| | | Oral hairy leukoplakia | 10030979 | |
| Parasites | Trypanosoma cruzi | None | | Narrow |
| | infection (Chagas'<br>Disease) (disseminated | American<br>trypanosomiasis | 10001935 | Broad |
| | disease only) (V) | Trypanosomiasis | 10044707 | |
| | | Meningitis<br>trypanosomal | 10027258 | |
| | Cryptosporidium species (chronic disease only) | Biliary tract infection cryptosporidial | 10067319 | Narrow |
| | (IV) | Cryptosporidiosis infection | 10011502 | Broad |
| | | Gastroenteritis<br>cryptosporidial | 10017899 | |
| | Leishmaniasis (Visceral | Visceral leishmaniasis | 10047505 | Narrow |
| | only) (IV) | Leishmaniasis | 10024198 | Broad |
| | Stronglyoides<br>(hyperinfection syndrome | None | | Narrow |
| | and disseminated forms only) (IV) | Strongyloidiasis | 10042254 | Broad |
| | Toxoplasmosis (IV) | Cerebral toxoplasmosis | 10057854 | Narrow |
| | | Eye infection toxoplasmal | 10015939 | |
| | | Hepatitis toxoplasmal | 10019798 | |
| | | Meningitis toxoplasmal | 10048848 | |
| | | Myocarditis toxoplasmal | 10028617 | |
| | | Pneumonia toxoplasmal | 10067566 | |
| | | Toxoplasma serology | 10050941 | Broad |
| | Non angelf - t | Toxoplasmosis | 10044272 | Name |
| | Non-specific terms | None | l | Narrow |

| | | Delftia acidovorans | 10081339 | |
|---|---|---|---|---|
| | | infection | MINESTER TOTAL | |
| | | Sphingomonas | 10081563 | 1 |
| | | paucimobilis | And the second s | |
| | | bacteraemia | | |
| | | Central nervous system | 10080100 | Broad |
| | | immune reconstitution | | CORPOR SAME A COLOCO |
| | | inflammatory response | | |
| | | Abscess fungal | 10000269 | ] |
| | | Alternaria infection | 10054207 | 1 |
| | 1 | Arthritis fungal | 10060966 | |
| | | Biliary tract infection | 10065203 | 1 |
| | | fungal | | |
| | 1 | Central nervous system | 10072805 | 1 |
| | | fungal infection | | |
| | | Cerebral fungal | 10049657 | |
| | | infection | | ] |
| | | Encephalitis fungal | 10065170 | ] |
| | | Erythema induratum | 10015213 | |
| | | Eye infection fungal | 10015933 | |
| | | Fungaemia | 10017523 | |
| | | Fungal abscess central | 10017524 | |
| | | nervous system | | |
| Non-specific | | Fungal endocarditis | 10017529 | |
| terms | | Fungal labyrinthitis | 10065174 | |
| | | Fungal oesophagitis | 10049656 | |
| | | Fungal peritonitis | 10061138 | |
| | | Fungal pharyngitis | 10076516 | |
| | | Fungal retinitis | 10068613 | |
| | | Fungal sepsis | 10058872 | |
| | | Fungal urethritis | 10081163 | |
| | | Hepatic infection fungal | 10065217 | |
| | | Meningitis fungal | 10027236 | |
| | | Mycotic | 10063202 | |
| | | endophthalmitis | | |
| | | Myocarditis mycotic | 10059026 | |
| | | Oral fungal infection | 10061324 | ] |
| | | Oropharyngitis fungal | 10061891 | |
| | | Osteomyelitis fungal | 10065239 | ] |
| | | Otitis media fungal | 10065175 | ] |
| | | Pancreatitis fungal | 10065190 | ] |
| | | Pericarditis fungal | 10065220 | ] |
| | | Phaehyphomycosis | 10034799 | ] |
| | | Pneumonia fungal | 10061354 | ] |
| | | Pulmonary mycosis | 10037422 | ] |
| | | Pulmonary | 10068184 | |
| | | trichosporonosis | | ] |
| | | Sinusitis fungal | 10058678 | |

| | | Splenic infection fungal | 10065194 | 13 |
|---|---|---|---|---|
| | | Systemic mycosis | 10052366 | , |
| Pneumonia | Infective Pneumonia<br>SMQ | All PTs (exclude<br>COVID-19 and<br>influenza PTs) | 20000231 | Narrow |

Abbreviations: DNA = deoxyribonucleic acid; EBV= Epstein-Barr virus; HBV = hepatitis B virus; MedDRA = Medical Dictionary for Regulatory Activities; POI = potential opportunistic infections; PT = Preferred Term; PVAN = Polyomavirus-associated nephropathy; SMQ = Standardized MedDRA Query.

## 6.10. Appendix 10: List of Planned Laboratory Analytes with Reference Range Sources

Table APP.10.1. Planned Laboratory Analytes with Reference Range Sources

| Laboratory | Laboratory Analyte | Reference | Analy | ysis Type |
|---|---|---|---|---|
| Group/Order | | Range Name | Central | Outlier/Shift |
| | | | Tendency | Analysis |
| Hematology | | | | |
| 1 | Hemoglobin | LCTPB | Yes | Yes |
| 2 | Hematocrit | LCTPB | Yes | Yes |
| 3 | Erythrocyte Count | LCTPB | Yes | Yes |
| 4 | Mean Cell Volume | LCTPB | Yes | Yes |
| 5 | Mean Cell Hemoglobin | LCTPB | Yes | Yes |
| 6 | MCHC | LCTPB | Yes | Yes |
| 7 | Platelets | LCTPB | Yes | Yes |
| 8 | Leukocyte Count | LCTPB | Yes | Yes |
| 9 | Bands | LCTPB | Yes | Yes |
| 10 | Neutrophils | LCTPB | Yes | Yes |
| 11 | Lymphocytes | LCTPB | Yes | Yes |
| 12 | Monocytes | LCTPB | Yes | Yes |
| 13 | Eosinophils | LCTPB | Yes | Yes |
| 14 | Basophils | LCTPB | Yes | Yes |
| Chemistry | | protection of the second secon | 0000000 | School and |
| 1 | ALT/SGPT | Covance | Yes | Yes |
| 2 | AST/SGOT | Covance | Yes | Yes |
| 3 | Alkaline Phosphatase | Covance | Yes | Yes |
| 4 | Total Bilirubin | Covance | Yes | Yes |
| 5 | Direct Bilirubin | Covance | Yes | Yes |
| 6 | Albumin | LCTPB | Yes | Yes |
| 7 | Creatine Phosphokinase | LCTPB | Yes | Yes |
| 8 | Creatinine | Covance | Yes | Yes |
| 9 | Urea Nitrogen | LCTPB | Yes | Yes |
| 11 | estimated GFR | Covance | Yes | Yes |
| 12 | Creatinine Clearance | Covance | Yes | Yes |
| 13 | Sodium | LCTPB | Yes | Yes |
| 14 | Potassium | LCTPB | Yes | Yes |
| 15 | Calcium | LCTPB | Yes | Yes |
| 16 | Total Protein | LCTPB | Yes | Yes |
| 17 | Fasting Glucose | LCTPB | Yes | Yes |
| 18 | Glucose, Non-Fasting or Random | LCTPB | Yes | Yes |
| 19 | Uric Acid | LCTPB | Yes | Yes |
| 20 | Cholesterol | LCTPB | Yes | Yes |
| 21 | Triglycerides | LCTPB | Yes | Yes |
| 22 | LDL Cholesterol – Direct | Covance | Yes | Yes |
| 23 | HDL Cholesterol – Direct | Covance | Yes | Yes |
| 24 | LDL/HDL Ratio – Calculated | None | Yes | No |

| Laboratory | Laboratory Analyte | Reference | | ysis Type |
|---|---|---|---|---|
| Group/Order | | Range Name | Central | Outlier/Shift |
| | | | Tendency | Analysis |
| Immunoglobu | lins | | | 200.00 |
| 1 | Immunoglobulin A | Covance | Yes | Yes |
| 2 | Immunoglobulin G | Covance | Yes | Yes |
| 3 | Immunoglobulin M | Covance | Yes | Yes |
| Urinalysis | | | | |
| 1 | Specific Gravity | LCTPB | Yes | Yes |
| 2 | pH | LCTPB | Yes | Yes |
| 3 | UA-color | None | No | Yes |
| 4 | UA-glucose | None | No | Yes |
| 5 | UA-protein | None | No | Yes |
| 6 | UA-bilirubin | None | No | Yes |
| 7 | UA-urobilinogen | None | No | Yes |
| 8 | UA-nitrites | None | No | Yes |
| 9 | UA-leukoesterase | None | No | Yes |
| 10 | UA-ketones | None | No | Yes |
| 11 | UA-occult blood | None | No | Yes |
| Flow Cytomet | | | 507 | |
| 1 | CD3+ T Cells – % | Covance | Yes | Yes |
| 2 | CD3+ T Cells – Absolute | Covance | Yes | Yes |
| 3 | CD3+CD4+ T cells (CD4) – % | Covance | Yes | Yes |
| 4 | CD3+CD4+ T cells (CD4) – | Covance | Yes | Yes |
| • | Absolute | Covance | 103 | 163 |
| 5 | CD3+CD8+ T cells (CD8) – % | Covance | Yes | Yes |
| 6 | CD3+CD8+ T cells (CD8) - 70 | Covance | Yes | Yes |
| O | Absolute | Covance | 103 | 103 |
| 7 | CD56+/CD16+ NK cells – % | Covance | Yes | Yes |
| 8 | CD56+/CD16+ NK cells – Absolute | Covance | Yes | Yes |
| 9 | CD19+ B cells – % | Covance | Yes | Yes |
| 10 | CD19+ B cells – 96<br>CD19+ B cells – Absolute | Covance | | Yes |
| 11 | CD4+CXCR3+CCR6- Th1 cells - % | None | Yes | |
| | | | Yes | No |
| 12 | CD4+CXCR3+CCR6- Th1 cells - | None | Yes | No |
| 12 | Absolute | N | 37 | NT |
| 13 | CD4+CXCR3-CCR6+ Th17 cells - | None | Yes | No |
| 14 | % CD4+CXCR3-CCR6+ Th17 cells - | None | Vas | No |
| 14 | Absolute | None | Yes | No |
| 15 | CD3+CD4+CD127- | Nama | Vac | NT |
| 13 | | None | Yes | No |
| | /loCD25+FoxP3+ (CD4+) T | | | |
| 1.0 | regulatory cells - % | ** | ** | 3.7 |
| 16 | CD3+CD4+CD127- | None | Yes | No |
| | /loCD25+FoxP3+ (CD4+) T | | | |
| | regulatory cells - Absolute | | | |
| 17 | CD3+CD4+CD127-/loCD25+ | None | Yes | No |
| | (CD4+) IL2-producing naïve and | | | |
| | central memory Helper T cells - | | | |
| | % | | | |

| Laboratory | Laboratory Analyte | Reference | Analysis Type | |
|---|---|---|---|---|
| Group/Order | | Range Name | Central Outlier/Shi | |
| | | | Tendency | Analysis |
| 18 | CD3+CD4+CD127-/loCD25+ | None | Yes | No |
| | (CD4+) IL2-producing naïve and | | | |
| | central memory Helper T cells - | | | |
| | Absolute | | | |
| 19 | CD20+ B cells – % | None | Yes | No |
| 20 | CD20+ B cells – Absolute | None | Yes | No |
| 21 | CD19+CD27-IgD+ mature naïve | None | Yes | No |
| | B cells – % | | | |
| 22 | CD19+CD27-IgD+ mature naïve | None | Yes | No |
| | B cells – Absolute | | | |
| 23 | CD19+CD27+IgD- switched | None | Yes | No |
| | memory B cells - % | | | |
| 24 | CD19+CD27+IgD- switched | None | Yes | No |
| | memory B - Absolute | | | |
| 25 | CD19+CD27+IgD+ non-switched | None | Yes | No |
| | memory B cells – % | | | |
| 26 | CD19+CD27+IgD+ non-switched | None | Yes | No |
| | memory B – Absolute | | | |
| 27 | CD19+CD27-IgD- | None | Yes | No |
| | Immature/transitional B cells - % | | | |
| 28 | CD19+CD27-IgD- | None | Yes | No |
| | Immature/transitional B - | | | |
| | Absolute | | | |
| 29 | CD4/CD8 Ratio - Calculated | None | Yes | No |
| | CD4+CD45RA-CCR7- effector | None | No | No |
| | memory T cells | | | |
| | CD4+CD45RA+CCR7- effector | None | No | No |
| | memory T cells | 5,15,755, | 50.50 | -1- |
| | CD4+CD45RA+CCR7- naïve T | None | No | No |
| | cells | = 1.Hent. | .m.v.m.v | #.X#X |
| : | CD4+CD45RA-CCR7+ central | None | No | No |
| | memory T cells | | | - 100 |
| | CD8+CD45RA+CCR7+ naïve T | None | No | No |
| | cells | 110110 | 110 | 1,0 |
| | CD8+CD45RA-CCR7+ central | None | No | No |
| | memory T cells | | | 2.0 |
| | CD8+CD45RA-CCR7- effector | None | No | No |
| | memory T cells | distribute. | - 10 | 410 |
| : | CD8+CD45RA+CCR7- effector | None | No | No |
| | memory T cells | 1,000 | 2.130 | 110 |

Abbreviations: ALT/SGPT = alanine aminotransferase/serum glutamic pyruvic transaminase;

AST/SGOT = aspartate aminotransferase/serum glutamic oxaloacetic transaminase; CD = cluster of differentiation; eGFR = estimated glomerular filtration rate; HDL = high-density lipoprotein;

Ig = immunoglobulin; IL = interleukin; LCTPB = Lilly Large Clinical Trial Population Based;

LDL = low-density lipoprotein; MCHC = mean corpuscular hemoglobin concentration; NK = natural killer; Th cells = Helper T cells; UA = urinalysis.

## 6.11. Appendix 11: Common Terminology Criteria for Adverse Events Related to Myelosuppressive Events

Table APP.11.1. CTCAE Related to Myelosuppressive Events

| _ | Laboratory | | Criteria in Système | Criteria in Conventional |
|---|---|---|---|---|
| Event | Test | Grade | International (SI) Units | (CN) Units |
| Anemia <sup>a</sup> | Hemoglobin | 0 | ≥7.27 mmol (Fe)/L for | ≥12 g/dL for females and |
| | | (normal) | females and ≥8.18 mmol | ≥13.5 g/dL for males |
| | | | (Fe)/L for males | |
| | | 1 | <7.27 mmol (Fe)/L for | <12 g/dL for females and |
| | | | females and 8.18 mmol | 13.5 g/dL for males and |
| | | | (Fe)/L for males and ≥6.2 | ≥10 g/dL |
| | | | mmol (Fe)/L | |
| | | 2 | <6.2 mmol (Fe)/L and ≥4.9 | <10 g/dL and ≥8.0 g/dL |
| | | | mmol (Fe)/L | |
| | | 3 | <4.9 mmol (Fe)/L and ≥4.0 | $<$ 8.0 g/dL and $\ge$ 6.5 g/dL |
| | | | mmol (Fe)/L | |
| EVANOR BENEFIT OF STREET | | 4 | <4.0 mmol (Fe)/L | <6.5 g/dL |
| Leukopenia <sup>a</sup> | White blood | 0 | ≥4.0 billion cells/L | ≥4.0 thousand cells/uL |
| | cell (WBC) | (normal) | | |
| | count | 1 | <4.0 billion cells/L and ≥3.0 | <4.0 thousand cells/uL and |
| | | | billion cells/L | ≥3.0 thousand cells/uL |
| | | 2 | <3.0 billion cells/L and ≥2.0 | <3.0 thousand cells/uL and |
| | | 124 | billion cells/L | ≥2.0 thousand cells/uL |
| | | 3 | <2.0 billion cells/L and ≥1.0 | <2.0 thousand cells/uL and |
| | | | billion cells/L | ≥1.0 thousand cells/uL |
| wasto or displayed | 974a - 50 - 77 | 4 | <1.0 billion cells/L | <1.0 thousand cells/uL |
| Neutropeniaa | Absolute | 0 | ≥2 billion cells/L | ≥2 thousand cells/uL |
| | neutrophil | (normal) | | - 9 |
| | count | 1 | <2 billion cells/L and ≥1.5 | <2 thousand cells/uL and |
| | (ANC) | No. | billion cells/L | ≥1.5 thousand cells/uL |
| | | 2 | <1.5 billion cells/L and ≥1.0 | <1.5 thousand cells/uL and |
| | | | billion cells/L | ≥1.0 thousand cells/uL |
| | | 3 | <1.0 billion cells/L and ≥0.5 | <1.0 thousand cells/uL and |
| | | | billion cells/L | ≥0.5 thousand cells/uL |
| SE SECTION SECURIS | William Baran W. | 4 | <0.5 billion cells/L | <0.5 thousand cells/uL |
| Lymphopenia <sup>a</sup> | Lymphocyte | 0 | ≥1.1 billion cells/L | ≥1.1 thousand cells/uL |
| | count | (normal) | | |
| | | 1 | <1.1 billion cells/L and ≥0.8 | <1.1 thousand cells/uL and |
| | | | billion cells/L | ≥0.8 thousand cells/uL |
| | | 2 | <0.8 billion cells/L and ≥0.5 | <0.8 thousand cells/uL and |
| | | | billion cells/L | ≥0.5 thousand cells/uL |
| | | 3 | <0.5 billion cells/L and ≥0.2 | <0.5 thousand cells/uL and |
| | | | billion cells/L | ≥0.2 thousand cells/uL |
| | | | <0.2 billion cells/L | ≥0.2 mousand cens/ull |

| Event | Laboratory<br>Test | Grade | Criteria in Système<br>International (SI) Units | Criteria in Conventional (CN) Units |
|---|---|---|---|---|
| Thrombocytopenia <sup>a</sup> | Platelet | 0 | ≥150 billions/L | ≥150 thousands/uL |
| | count | (normal) | | |
| | | 1 | <150 billions/L and ≥75 billions/L | <150 thousands/uL and ≥75 thousands/uL |
| | | 2 | <75 billions/L and ≥50 billions/L | <75 thousands/uL and ≥50 thousands/uL |
| | | 3 | <50 billions/L and ≥25 billions/L | <50 thousands/uL and ≥25 thousands/uL |
| | | 4 | <25 billions/L | <25 thousands/uL |

Abbreviations: CTCAE = Common Terminology Criteria for Adverse Events; Fe = iron.

a CTCAE grading was adjusted by replacing lower limit of normal with a single value.

## Signature Page for VV-CLIN-117498 v1.0

| Approval | PPD |
|----------|-------------------------------|
| | 31-Aug-2023 15:54:53 GMT+0000 |

Signature Page for VV-CLIN-117498 v1.0